BI Study Number: 1237.51

## SATisfaction and adherence to COPD treatment

## STATISTICAL ANALYSIS PLAN

Version 1.5, 22/09/2017

| Written by | |
|-------------|--------------------------------------|
| Role | Biostatistician |
| Date | |
| Signature | |
| Reviewed by | |
| Role | Data Management &<br>Statistics Unit |
| Date | |
| Signature | |



## **INDEX**

| LIS' | OF ABBREVIATIONS | |
|---|---|---|
| | STATISTICAL AANALYSIS PLAN OBJECTIVES | 6 |
| 2 | DEFINITION OF EVALUABLE PATIENTS | 7 |
| 3 | COMPUTED VARIABLES | |
| ĺ | CONTENTS | |
| · | 1 Patient disposition | |
| 7 | Table 1. Enrolled and evaluable patients | |
| | Table 2. Reasons for non-eligibility to analyses | |
| | Table 3. Premature study termination | |
| 4 | 2 Demographics and baseline characteristics | |
| | Table 4. Socio-demographic characteristics at enrollment | 10 |
| | Table 5. Smoke habilts at enrollment | |
| | Table 6. COPD medical history at enrollment | |
| | Table 7. Comorbidities at enrollment. | |
| | Table 8. Vital signs at enrollment | |
| | Table 9. Respiratory Functions at enrollment | |
| 4 | 3 Patients' satisfaction for medical treatment (TSQM-9) (primary objective) | |
| | Table 10. Patients' satisfaction for medical treatment (TSQM-9 items) at each study visit | |
| | Table 11. Patients' satisfaction for medical treatment (TSQM-9 subscales) at each study visit | |
| 4 | 4 Patients' disease perception (B-IPQ) (secondary objective #1) | |
| | Table 12. Patients' disease perception (B-IPQ) at each study visit | |
| 4 | 5 Patients' adherence to COPD treatment (MMAS-4) (secondary objective #1) | |
| | Table 13. Patients' adherence to COPD treatment (MMAS-4) at each study visit | |
| 4 | 6 Patients' health status (CAT) (secondary objective #1) | |
| | Table 14. Patients' health status (CAT) at each study visit | 21 |
| 4 | 7 Patients' dyspnea (mMRC) (secondary objective #1) | 22 |
| | Table 15. Patients' dyspnea (mMRC) at each study visit | |
| 4 | 8 Patients' COPD awareness | |
| | Table 16. Patients' COPD awareness (Awareness structured interview) each study visit | |
| | 9 Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period | |
| ( | secondary objective #2) | 23 |
| | Table 17. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation per | |
| | (Repeated measures regression models) – Effectiveness domain | 23 |
| | (Repeated measures regression models) – Convenience domain | |
| | Table 19. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation per | |
| | (Repeated measures regression models) – Global satisfaction domain | |
| 4 | 10 Healthcare resource utilization (secondary objective #3) | |
| - 7 | Table 20. Hospitalizations not in ICU during observation period: patients' distribution | |
| | Table 21. Hospitalizations not in ICU during observation period: details | |
| | Table 22. Hospitalizations in ICU during observation period: patients' distribution | |
| | Table 23. Hospitalizations in ICU during observation period: details | |
| | Table 24. Emergency room accesses: patients' distribution | |
| | Table 25. Emergency room accesses: details | |
| | Table 26. Specialist outpatient visits: patients' distribution. | |
| | Table 27. General practitioner visits: patients' distribution | |
| | Table 28. Laboratory tests: patients' distribution | |
| | Table 29. Laboratory tests: details. | |
| | Table 30. Oxygen therapy | |
| | Table 31. List of oxygen therapies | |
| | Table 32. Patients receiving fixed/non-fixed dose therapies for COPD at enrollment | |
| | Table 33. COPD pharmacological treatments ongoing at enrollment | |
| | Table 34. COPD pharmacological treatments ongoing at 6-month follow-up visit | |
| | Table 35. COPD pharmacological treatments ongoing at 12-month follow-up visit | |
| | Table 36 Medications for adverse events | 26 |

| | 4.11 | Correlation between patients' satisfaction and resource utilization (secondary objective #4) | |
|---|---|---|---|
| | Table | 37. Correlation between patients' satisfaction and resource utilization (including drugs) | |
| | 4.12 | Exacerbations | 27 |
| | Table | 38. Exacerbations: patients' distribution | 27 |
| | Table | 39. Exacerbations: details | 27 |
| | 4.13 | Safety | 28 |
| | Table | 40. Overall Summary of Adverse Events and Adverse Event Reactions | |
| | | able will provide: | |
| | | 41. Patients' distribution by type of adverse event | |
| | | 42. Distribution of type of adverse event: details. | |
| | | 43. List of adverse events | |
| | | 44. Pregnancies: patients' distribution. | |
| | 4.14 | Supportive analysis | |
| | | 45. Patients' satisfaction for medical treatment (TSQM-9 items) at each study visit - Switchers vs non-switchers | |
| | | 46. Patients' satisfaction for medical treatment (TSQM-9 subscales) at each study visit- Switchers vs non-switchers | |
| 5 | | LES LAYOUT. | |
| , | 5.1 | Patient disposition | |
| | | 1. Enrolled and evaluable patients | |
| | | Reasons for non-eligibility to analyses | |
| | | Reasons for non-eligibility to analyses Premature study termination | |
| | 5.2 | Demographics and baseline characteristics. | |
| | | 4. Socio-demographic characteristics at enrollment | |
| | | Socio-demographic characteristics at enrollment. Smoke habilts at enrollment | |
| | | Smoke nabilits at enrollment COPD medical history at enrollment | |
| | | 7. Comorbidities at enrollment | |
| | | 8. Vital signs at enrollment | |
| | | 9. Respiratory Functions at enrollment | |
| | 5.3 | Patients' satisfaction for medical treatment (TSQM-9) (primary objective) | |
| | | 10. Patients' satisfaction for medical treatment (TSQM-9 items) at each study visit | |
| | | 11. Patients' satisfaction for medical treatment (TSQM-9 subscales) at each study visit | |
| | 5.4 | Patients' disease perception (B-IPQ) (secondary objective #1) | |
| | | 12. Patients' disease perception (B-IPQ) at each study visit | |
| | 5.5 | Patients' adherence to COPD treatment (MMAS-4) (secondary objective #1) | |
| | | 13. Patients' adherence to COPD treatment (MMAS-4) at each study visit | |
| | 5.6 | Patients' health status (CAT) (secondary objective #1) | |
| | | 14. Patients' health status (CAT) at each study visit | |
| | 5.7 | Patients' dyspnea (mMRC) (secondary objective #1) | |
| | | 15. Patients' dyspnea (mMRC) at each study visit | |
| | 5.8 | Patients' COPD awareness | |
| | | 16. Patients' COPD awareness (Awareness structured interview) each study visit | 45 |
| | 5.9 | Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period | 40 |
| | (seconda | ary objective #2) | 48 |
| | | 17. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period | |
| | (Repe | eated measures regression models) – Effectiveness domain | 48 |
| | rable | 18. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period | )a |
| | (Repe | eated measures regression models) – Convenience domain | 48 |
| | | 19. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period | |
| | | eated measures regression models) – Global satisfaction domain | |
| | 5.10 | Healthcare resource utilization (secondary objective #3) | |
| | | 20. Hospitalizations not in ICU during observation period: patients' distribution | |
| | | 21. Hospitalizations not in ICU during observation period: details | |
| | | 22. Hospitalizations in ICU during observation period: patients' distribution | |
| | | 23. Hospitalizations in ICU during observation period: details | |
| | | 24. Emergency room accesses: patients' distribution | |
| | | 25. Emergency room accesses: details | |
| | | 26. Specialist outpatient visits: patients' distribution. | |
| | | 27. General practitioner visits: patients' distribution | |
| | l able | 28. Laboratory tests: patients' distribution | 54 |

| | Table | 29. Laboratory tests: details | . 54 |
|---|---|---|---|
| | Table | 30. Oxygen therapy | . 55 |
| | Table | 31. List of oxygen therapies | . 55 |
| | | 32. Patients receiving fixed/non-fixed dose therapies for COPD at enrollment | |
| | | 33. COPD pharmacological treatments ongoing at enrollment | |
| | | 34. COPD pharmacological treatments ongoing at 6-month follow-up visit | |
| | | 35. COPD pharmacological treatments ongoing at 12-month follow-up visit | |
| | | 36. Medications for adverse events | |
| | 5.11 | Correlation between patients' satisfaction and resource utilization (secondary objective #4) | . 57 |
| | Table | 37. Correlation between patients' satisfaction and resource utilization (including drugs) | |
| | 5.12 | Exacerbations | |
| | Table | 38. Exacerbations: patients' distribution | . 58 |
| | | 39. Exacerbations: details | |
| | 5.13 | Safety | . 59 |
| | Table | 40. Overall Summary of Adverse Events and Adverse Event Reactions | . 59 |
| | | 41. Patients' distribution by type of adverse event | |
| | | 42. Distribution of type of adverse event: details | |
| | | 43. List of adverse events | |
| | Table | 44. Pregnancies: patients' distribution | . 61 |
| | 5.14 | Supportive analysis | |
| | Table | 45. Patients' satisfaction for medical treatment (TSQM-9 items) at each study visit - Switchers vs non-switchers | . 61 |
| | Table | 46. Patients' satisfaction for medical treatment (TSQM-9 subscales) at each study visit- Switchers vs non-switchers | . 61 |
| 6 | QUA | LITY CHECKS ON THE STATISTICAL REPORT | <b>62</b> |
| 7 | REVI | SION HISTORY | 64 |
| 2 | | NDICES | |
| | 8.1 | COPD awareness questionnaire scoring system | |
| | 8.2 | Modified Medical Research Council (mMRC) dyspnoea scale | |
| | 8.3 | Treatment Satisfaction Questionnaire for Medication (TSQM-9) | |
| | 8.4 | COPD Assessment Test (CAT) | |
| | 8.5 | Brief Illness Perception Questionnaire (B-IPQ) | |
| | 8.6 | Morisky Medication Adherence Scale (MMAS-4) | 76 |

#### LIST OF ABBREVIATIONS

ACOS Asthma COPD Overlap Syndrome

ADR Adverse Drug Reaction

AE Adverse Event

BI Boheringer Ingelheim Italy S.p.A
B-IPQ Brief-Illness Perception Questionnaire

BMI Body Mass Index BS Biostatistician

CAT COPD Assessment Test CDM Clinical Data Manager

COPD Chronic Obstructive Pulmonary Disease
DLCO Diffusion Lung Capacity for carbon monoxide

eCRF electronic Case Report Form

ER Emergency Room FAS Full Analysis Set

FEV1 Forced Expiratory Volume in the 1st second

FVC Forced Vital Capacity
ICS Inhaled corticosteroids
ICU Intensive Care Unit
LABA Long-acting β2-agonists

LAMA Long-acting muscarinic agonists

Max Maximum Min Minimum

MMAS-4 Morisky medication Adherence Scale, 4 items mMRC modified Medical Research Council dyspnea scale

N Number of observations

NA Not Available NK Not Known

PDE4-I Phosphodiesterase type 4 inhibitors

PRO Patient-Reported Outcome

R-DMS Responsible Data Management and Statistics Unit

SABA Short-acting β-agonists SAE Serious Adverse Event

SAMA Short-acting muscarinic agonists

SAP Statistical Analysis Plan SD Standard Deviation TLC Total Lung Capacity

TSQM-9 Treatment Satisfaction Questionnaire for Medication, 9 items

VC Vital Capacity

#### 1 STATISTICAL AANALYSIS PLAN OBJECTIVES

The SATisfaction and adherence to COPD treatment study (i.e. SAT study) is a multi-center, non-interventional (observational) cohort study based mainly on newly collected data. About 400 consecutive COPD patients will be enrolled in approximately 8 months (from first patient enrolled). Patients will be followed up for 1 year, with an intermediate evaluation after 6 (+/-1) months from baseline (which is compatible with current clinical practice in Italy for COPD patients management).

The present Statistical Analysis Plan has beed designed considering the following input documents:

- the Study Protocol v.1.0 31/07/2015,
- the electronic case report form v. 1.2 27/04/2016;
- the minutes of the Customer's Meeting held on the 26/06/2017.

This SAP is aimed at evaluating the following SAT study objectives:

## Primary objective:

To describe the patients' satisfaction to COPD medical treatments (by means of the TSQM9) during a 12-month observation period (namely, at enrolment, and after 6 and 12 months) in real- world setting.

## Secondary objectives:

- To describe patient disease perception (by means of illness perception questionnaire B-IPQ), adherence to COPD treatment (by means of MMAS4), health status (by means of CAT questionnaire) and dyspnea (by means of mMRC) during a 12-month observation period.
- 2. To analyze the relation between treatment satisfaction and demographic (such as age, gender), clinical (such as number of exacerbations, spirometric parameters) parameters and PROs during a 12-month observation period.
- 3. To describe the health care resources utilization and related cost according to the Italian National Health Service (INHS) during a 12-month observation period.
- 4. To assess the correlation between patients' satisfaction and resource utilization.

In this document the eCRF fields are indicated as follows: "label of the field" [name of the eCRF form.name of the variable in the dataset].

## 2 DEFINITION OF EVALUABLE PATIENTS

## 2.1 Patients evaluable at enrolment (FULL ANALYSIS SET)

All enrolled patients meeting the following inclusion / exclusion / other criteria listed in the present paragraph will be considered evaluable at enrollment (Full analysis set) (i.e. COPD patients aged ≥40 years, with stable pharmacological treatment for COPD and no exacerbations for at least 3 months, who signed informed consent and privacy form, with at least one Treatment Satisfaction Questionnaire for Medication (TSQM-9) domain score calculated at enrollment visit):

#### Inclusion criteria

Criterion 1: Patients aged ≥40 years

- Question "1. Is the patient aged ≥40 years?" = "Yes" [F01\_INC\_EXC\_CRITERIA.CI\_1] AND
- Inclusion criterion "1. Patients aged ≥40 years?" not checked in the PROTOCOL DEVIATION FORM.
   [F24\_PROTOCOL\_DEVIATION\_FORM. PD\_CI\_1] AND
- Age at enrollment visit (years) ≥ 40 [\_PatientInfo.Age]

Criterion 2: Patients must have a documented diagnosis of chronic obstructive pulmonary disease (COPD)

- Question "2. Has the patient a documented diagnosis of chronic obstructive pulmonary disease (COPD)?" =
   "Yes" [F01\_INC\_EXC\_CRITERIA.CI\_2]
   AND
- Inclusion criterion "2. Patients must have a documented diagnosis of chronic obstructive pulmonary disease (COPD)" not checked in the PROTOCOL DEVIATION FORM [F24\_PROTOCOL\_DEVIATION\_FORM.
   PD CI 2] AND
- Date of COPD diagnosis (mm/yyyy) not missing [F04\_COPD\_MEDICAL\_HISTORY.MH\_Date\_diagnosis]

Criterion 3: Patients with no exacerbations in the last 3 months

- Question "3. Patient without any exacerbation in the last 3 months" = "Yes"
   [F01\_INC\_EXC\_CRITERIA.QUESTION 3. CI\_3] AND
- Inclusion criterion "3. Patients with no exacerbations in the last 3 months" not checked in the PROTOCOL DEVIATION FORM [F24\_PROTOCOL\_DEVIATION\_FORM. PD\_CI\_3] AND
- Onset dates at each follow-up visit (Row 1 to 10) [F08\_EXACERBATIONS.Ex\_exacer\_1-10\_onset\_date] >
   Date of enrolment visit (dd/mm/yyyy) [\_PatientInfo.Date\_enrollment]

Criterion 4: Patients requiring regular treatment according to GOLD guidelines, i.e.: undergoing stable pharmacological treatment for COPD since at least 3 months

- Question "4. Does the patient require a regular treatment according to GOLD guidelines, i.e.: undergoing stable pharmacological treatment for COPD since at least 3 months?" = "Yes" [F01\_INC\_EXC\_CRITERIA.CI\_4] AND
- Inclusion criterion "4. Patients requiring regular treatment according to GOLD guidelines, i.e.: undergoing stable pharmacological treatment for COPD since at least 3 months" not checked in the PROTOCOL DEVIATION FORM [F24 PROTOCOL DEVIATION FORM. PD\_CI\_4] AND
- COPD Pharmacological therapy form: Start date of therapy (dd/mmm/yyyy) not missing AND (Start date of therapy (dd/mmm/yyyy) [F20\_COPD PHARMACOLOGICAL THERAPY.START\_DATE\_THER] < Date of enrolment visit (dd/mm/yyyy) 3\*30.4375 [\_PatientInfo.Date\_enrollment] OR Start date of therapy (dd/mmm/yyyy) > Date of enrolment visit (dd/mm/yyyy)) AND
- COPD Pharmacological therapy form: End date of therapy (dd/mmm/yyyy) [F20\_COPD PHARMACOLOGICAL THERAPY.END\_DATE\_THER] = missing OR End date of therapy (dd/mmm/yyyy) > Date of enrolment visit (dd/mm/yyyy) [\_PatientInfo.Date\_enrollment]

Criterion 5: Written informed consent to both participation in the study and privacy form

- Question "5. Is a written informed consent to both participation in the study and privacy form available?" =
   "Yes" [F01\_INC\_EXC\_CRITERIA.CI\_5] AND
- Inclusion criterion "5. Written informed consent to both participation in the study and privacy form" not checked in the PROTOCOL DEVIATION FORM [F24\_PROTOCOL\_DEVIATION\_FORM. PD\_CI\_5] AND
- Date of informed consent signature (dd/mm/yyyy) not missing [\_PatientInfo.Date\_CI] AND
- Date of privacy form signature (dd/mm/yyyy) not missing [\_PatientInfo.Date\_privacy] AND
- Date of informed consent signature (dd/mm/yyyy) = Date of privacy form signature (dd/mm/yyyy) AND
- Date of informed consent signature (dd/mm/yyyy) ≤ Date of enrolment visit (dd/mm/yyyy)

Criterion 6: Patients capable of discernment and able to read or write in Italian language

- Question "6. Is the patient capable of discernment and able to read or write in Italian language?" = "Yes"
   [F01 INC EXC CRITERIA.CI 6] AND
- Inclusion criterion "6. Patients capable of discernment and able to read or write in Italian language" not checked in the PROTOCOL DEVIATION FORM [F24\_PROTOCOL\_DEVIATION\_FORM. PD\_IC\_6]

### Exclusion criteria

Criterion 7: Patients who are currently participating in a clinical trial on experimental drugs

- Question "7. Does the patient currently participate in a clinical trial on experimental drugs?" = "No"
   [F01\_INC\_EXC\_CRITERIA.EC\_1] AND
- Exclusion criterion "1. Patients who are currently participating in a clinical trial on experimental drugs" not checked in the PROTOCOL DEVIATION FORM [F24\_PROTOCOL\_DEVIATION\_FORM. PD\_EC\_1]

Criterion 8: Patients naïve to pharmacological treatment for COPD

- Question "8. Is the patient naïve to pharmacological treatment for COPD?" = "No"
   IF01 INC EXC CRITERIA.EC 21 AND
- COPD Pharmacological therapy form: Start date of therapy (dd/mmm/yyyy) (earliest record) not missing AND
- Exclusion criterion "2. Patients naïve to pharmacological treatment for COPD" not checked in the PROTOCOL DEVIATION FORM [F24 PROTOCOL DEVIATION FORM. PD EC 2]

Criterion 9: Diagnosis of Asthma COPD Overlap Syndrome (ACOS)

- Question "9. Does the patient have a diagnosis of Asthma COPD Overlap Syndrome (ACOS)? " = "No"
   [F01 INC EXC CRITERIA.EC 3] AND
- Exclusion criterion "3. Diagnosis of Asthma COPD Overlap Syndrome (ACOS)" not checked in the PROTOCOL DEVIATION FORM [F24 PROTOCOL DEVIATION FORM. PD\_EC\_3]

## Other criteria

Criterion 10: patients with at least one Treatment Satisfaction Questionnaire for Medication (TSQM-9) domain score calculated at enrollment visit

- TSQM-9 items #1,2,3 [TSQM9 1-3] not missing & ≠ "Non risponde" at enrollment visit, OR
- TSQM-9 items #4,5,6 [TSQM9\_4-6] not missing & ≠ "Non risponde" at enrollment visit, OR
- TSQM-9 items #7,8,9 [TSQM9\_7-9] not missing & ≠ "Non risponde" at enrollment visit

### 2.2 Patients evaluable at 6-month follow-up

All enrolled patients meeting the following criteria will be considered evaluable at enrollment and at 6 month follow-up visit:

Patients considered evaluable at enrollment (i.e., responding to criteria of par 2.1 Full Analysis Set) who fulfill also the following criteria (i.e. all FAS patients who performed the 6-month follow-up visit and with at least one Treatment Satisfaction Questionnaire for Medication (TSQM-9) domain score calculated at the 6-month follow-up visit).

Criterion 11: Data collected at 6-month follow-up

"Data collected at 6 (±1) month follow up?" = "Yes" [F19\_PATIENT\_DISPOSITION, 6 month f-up.PD\_1]

Criterion 12: Follow-up performed 6+/- 1 month from enrollment

- (Date of follow up visit (dd/mmm/yyyy) [F19\_PATIENT\_DISPOSITION, 6 month f-up.PD\_2] Date of enrolment visit (dd/mm/yyyy) [\_PatientInfo. Date\_enrollment]/30.4375 ≥ 5) AND
- (Date of follow up visit (dd/mmm/yyyy) [F19\_PATIENT\_DISPOSITION, 6 month f-up.PD\_2] Date of enrolment visit (dd/mm/yyyy) [\_PatientInfo. Date\_enrollment] /30.4375 ≤ 7)

The Biostatistician will evaluate the opportunity to apply a tolerance window during the analysis of data; the Sponsor will be informed of any possible changes in this range.

Criterion 13: patients with at least one Treatment Satisfaction Questionnaire for Medication (TSQM-9) domain score calculated at 6-month follow-up visit

- TSQM-9 items #1,2,3 [TSQM9\_1-3] not missing & ≠ "Non risponde" at 6-month follow-up, OR
- TSQM-9 items #4,5,6 [TSQM9\_4-6] not missing & ≠ "Non risponde" at 6-month follow-up, OR
- TSQM-9 items #7,8,9 [TSQM9\_7-9] not missing & ≠ "Non risponde" at 6-month follow-up

## 2.3 Patients evaluable at 12-month follow-up

All enrolled patients meeting the following criteria will be considered evaluable at enrollment and at 12 month follow-up visit:

Patients considered evaluable at enrollment (i.e., responding to criteria of par 2.1 Full Analysis Set) who fulfill also the following criteria (i.e. all FAS patients who performed the 12-month follow-up visit and with at least one Treatment Satisfaction Questionnaire for Medication (TSQM-9) domain score calculated at the 12-month follow-up visit).

Criterion 14: Data collected at 12-month follow-up

"Data collected at 12 (±1) month follow up?" = "Yes" [F19\_PATIENT\_DISPOSITION, 12 month f-up.PD\_1]

Criterion 15: Follow-up performed 12+/- 1 month from enrollment

- (Date of follow up visit (dd/mmm/yyyy) [F19\_PATIENT\_DISPOSITION, 12 month f-up.PD\_2] Date of enrolment visit (dd/mm/yyyy) [\_PatientInfo. Date\_enrollment]/30.4375 ≥ 11) AND
- (Date of follow up visit (dd/mmm/yyyy) [F19\_PATIENT\_DISPOSITION, 12 month f-up.PD\_2] Date of enrolment visit (dd/mm/yyyy) [\_PatientInfo. Date\_enrollment] /30.4375 ≤ 13)

The Biostatistician will evaluate the opportunity to apply a tolerance window during the analysis of data; the Sponsor will be informed of any possible changes in this range.

Criterion 16: patients with at least one Treatment Satisfaction Questionnaire for Medication (TSQM-9) domain score calculated at 12-month follow-up visit

- TSQM-9 items #1,2,3 [TSQM9\_1-3] not missing & ≠ "Non risponde" at 12-month follow-up, OR
- TSQM-9 items #4,5,6 [TSQM9\_4-6] not missing & ≠ "Non risponde" at 12-month follow-up, OR
- TSQM-9 items #7,8,9 [TSQM9 7-9] not missing & ≠ "Non risponde" at 12-month follow-up

Three sets of patients have been identified for the evaluation of SAT study objectives.

Chart 1 displays the analysis sets considered for the statistical analyses foreseen in the Study Protocol.

Chart 1: Sets of patients considered for each statistical analysis

| | Patients evaluable at enrollment | Patients evaluable at enrollment and at 6 | Patients evaluable at enrollment and at |
|---|---|---|---|
| | (FAS) | month follow-up | 12 month follow-up |
| Enrolled and evaluable patients | X | X | Χ |
| Main socio-demographics and life habits | Χ | | |
| (age, gender, race, education, employment | | | |
| status) at enrollment | | | |
| Medical history for COPD (number of | X | | |
| exacerbations in the 12 months prior to enrollment) | | | |
| Patients' satisfaction to COPD medical | X* | X* | X* |
| treatments (by means of the TSQM9) at | | | |
| each study visit | | | |
| Patient disease perception (by means of | X* | X* | X* |
| illness perception questionnaire B-IPQ) at | | | |
| each study visit | | | |
| Patient adherence to COPD treatment (by | X* | X* | X* |
| means of MMAS4) at each study visit | | | |
| Patient health status (by means of CAT | X* | X* | X* |
| questionnaire) at each study visit | 20 | 201 | 200 |
| Measurement of dyspnea (by means of | X* | X* | X* |
| mMRC) at each study visit | X* | V* | V* |
| Patient's COPD awareness (COPD | X | X* | X* |
| awareness questionnaire) at each study visit | | | |
| Relation between treatment satisfaction and | | | X |
| demographic (such as age, gender), clinical | | | ^ |
| (such as number of exacerbations, | | | |
| spirometric parameters) parameters and | | | |
| PROs during a 12-month observation period | | | |
| Description of health care resources | Χ | | |
| utilization and related cost according to the | | | |
| Italian National Health Service (INHS) | | | |
| during a 12-month observation period. | | | |
| To assess the correlation between patients' | | | Χ |
| satisfaction and resource utilization during a | | | |
| 12-month observation period | | | |
| Ongoing pharmacological and non- | Х | | |
| pharmacological treatments for COPD | | | |
| Exacerbations occurred during observation | X | | |
| period | | | |

<sup>\*</sup>Patients having PRO score computable at the visit will be considered for this analysis (i.e. PRO filled in at the visit and having a sufficient number of items recorded to allow score computation (PROs computation details are reported in Section 3. "Computed Variables")).

## 2.4 Safety set

All enrolled patients meeting the inclusion criteria #4 and #5 and not meeting the exclusion criteria #7, #8 and #9 (i.e. all enrolled subjects who provided informed consent to both participation in the study and privacy form, requiring regular treatment according to GOLD guidelines) will be included in the safety analysis.

#### 3 COMPUTED VARIABLES

The following variables will be computed as described below.

#### **BMI Classes**

Underweight: BMI [F05\_PHYSICAL\_EXAMINATION.PE\_BMI] < 18.5, normal weight: BMI 18.5-24.9, overweight: BMI 25-29.9, obese: BMI >= 30.

## Age at COPD diagnosis

Is calculated as the difference between age at enrollment visit (years) [\_PatientInfo.Age] and the difference between the date of enrollment [\_PatientInfo.Date\_enrollment] and the date of COPD diagnosis[F04\_COPD\_MEDICAL\_HISTORY.MH\_Date\_diagnosis]/365.25.

## Smoking duration at enrolment (years)

For patient who are current smokers by the time of enrolment ([F03\_LIFE\_HABITS.RF\_smoking] = "Current smoker"):

Smoking duration at enrolment = YEAR(Date of enrolment visit [\_PatientInfo.Date\_enrollment]) - Start year [F03\_LIFE\_HABITS.RF\_start\_year\_Num], if Start year and Date of enrolment visit are not missing.

For patient who are former smokers by the time of enrolment ([F03\_LIFE\_HABITS.RF\_smoking] = "Former smoker"):

Smoking duration at enrolment = Stop year [F03\_LIFE\_HABITS.RF\_stop\_year\_Num] - Start year [F03\_LIFE\_HABITS.RF\_Start\_year\_Num], if Stop year and Start year are not missing.

## COPD duration (years)

Is calculated as the difference between the date of enrollment [\_PatientInfo.Date\_enrollment] and the date of COPD diagnosis[F04\_COPD\_MEDICAL\_HISTORY.MH\_Date\_diagnosis]/365.25.

## **COPD** severity

In patients with FEV1/FVC at a certain visit [F07\_FUNCTIONAL\_ASSESSMENT. FA\_FEV1\_FVC] < 70%, the patient's COPD severity will be assessed according to the FEV1 of the predicted (%) value reported at each visit [F07\_FUNCTIONAL\_ASSESSMENT. FA\_FEV1\_predicted].

In particular, patients will be classified in the following ordinal groups:

- GOLD 1 (Mild): FEV1 of the predicted (%) ≥ 80%;
- GOLD 2 (Moderate): 50% ≤ FEV1 of the predicted (%) < 80%;</li>
- GOLD 3 (Severe): 30% ≤ FEV1 of the predicted (%) < 50%;</li>
- GOLD 4 (Very Severe): FEV1 of the predicted (%) < 30%.

Source: GLOBAL STRATEGY FOR THE DIAGNOSIS, MANAGEMENT, AND PREVENTION OF CHRONIC OBSTRUCTIVE PULMONARY DISEASE - UPDATED 2015.

## COPD awareness questionnaire composite scores (from the COPD awareness structured interview)

The questionnaire is designed to measure patient's COPD awareness assessing the patient's knowledge of the disease, acceptance of the disease, perception of the disease and symptoms, and awareness of the patient's need to be treated.

Each COPD awareness questionnaire's item can be answered by means of a 4-point categorical scale (ranging from "I definitely do not agree" to "I totally agree"). However, the answer options are ordinal and, since they represent different grades of agreement, these answer options can be converted in a 4-point scale ranging from 0 to 3, as described in Appendix 8.1.

The COPD awareness questionnaire composite scores will be computed (according to the algorithm validated in the SAT substudy) starting from the scores given to non-missing items [F12\_AWARENESS. AWARENESS\_01 – AWARENESS\_27], after having assigned the appropriate weight to each item, as described in Appendix 8.1. In particular, the following composite scores can be computed:

- 'Acknowledgement of disease' domain score (ranging from 0 to 15) is computed as the sum of the items #7,
   #15, #22, #24, and #25, when all of them are not missing;
- 'Awareness of treatment needs' domain score (ranging form 0 to 18) is computed as the sum of the items #4, #9, #12, #14, #18, and #23, when all of them are not missing;
- 'Knowledge of disease' domain score (ranging form 0 to 12) is computed as the sum of the items #1, #2, #19, and #26, when all of them are not missing;
- 'Disease perception' domain score (ranging form 0 to 15) is computed as the sum of the items #5, #8, #10, #20, and #21, when all of them are not missing;
- COPD awareness questionnaire total score (ranging form 0 to 60) is computed as the sum of all above-listed items, when all of them are not missing

Higher score reflect a patient's higher grade of awareness regarding his/her COPD in the respective investigated domain, and vice versa.

Changes in the COPD awareness questionnaire composite scores at each follow-up visit from enrollment will be calculated, for each patient, as the following difference: (composite score at 6/12 months - composite score at enrollment), if both scores are available.

## CAT score

The COPD Assessment Test (CAT) is an 8-item unidimensional measure of health status impairment in COPD (*P.W. Jones, G. Harding, P. Berry, I. Wiklund, W-H. Chen and N. Kline Leidy Development and first validation of the COPD Assessment Test. Eur Respir J 2009; 34: 648–654).* It is designed to measure the impact of COPD on a person's life, and how this changes over time. It contains eight short, simple, patient-completed questions. Patients can choose a score from 0 to 5 for the extent to which the described impairment is true for them, thereby providing a measure of the impact of COPD on their individual health.

The score ranges from 0 to 40; higher scores represent worse health.

The following categories can be identified on the basis of the CAT total score: < 10 : 10 - 20 : 21 - 30 : > 30.

The CAT score will be calculated as the sum of the responded items [F16 CAT.CAT ITEM 1 - CAT ITEM 8].

If more than two responses are missing, the score cannot be calculated; when one or two items are missing, their scores can be estimated by calculating the average of the non-missing item scores.

Changes in the CAT score at each follow-up visit from enrollment will be calculated, for each patient, as the following difference: (score at 6/12 months - score at enrollment), if both scores are available.

## B-IPQ total score

The Brief Illness Perception Questionnaire (B-IPQ) is a validated 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness (*Broadbent E et al. "The Brief Illness Perception Questionnaire"*. *Journal of Psychosomatic Research.* 2006; 60: 631–637). All of the questionnaire items (except the causal question, item 9) are rated using a 0-to-10 response scale. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5).

Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Assessment of the causal representation is by an opened response item, which asks patients to list the three most important causal factors in their illness (Item 9).

The B-IPQ total score will be computed as follows: the reversed scores of items 3, 4, and 7 [F14\_BIPQ.BIPQ\_3, BIPQ\_4, BIPQ\_7] will be added to the scores of items 1, 2, 5, 6, and 8 [F14\_BIPQ.BIPQ\_1, BIPQ\_2, BIPQ\_5, BIPQ\_6, BIPQ\_8]. A higher score reflects a more threatening view of the illness). The B-IPQ total score can be computed only if items #1-8 are filled in: only item 9 can be missing. Missing values will not be replaced.

Changes in the B-IPQ total score at each follow-up visit from enrollment will be calculated, for each patient, as the following difference: (score at 6/12 months - score at enrollment), if both scores are available.

#### TSQM-9 subscales scores

The Treatment Satisfaction Questionnaire for Medication, 9 items (TSQM-9) was derived from the original version, and it has a total of 9 items with responses to nearly all items rated on a five-point or seven-point rating scale that provide scores on three scales: effectiveness (3 items), convenience (3 items) and global satisfaction (3 items). The TSQM-9 domain scores (effectiveness, convenience and global satisfaction) will be calculated as recommended by the instrument authors (Atkinson MJ, Kumar R, Cappelleri JC, Hass SL: Hierarchical construct validity of the treatment satisfaction questionnaire for medication (TSQM version II) among outpatient pharmacy consumers. Value Health. 2005 Nov-Dec;8 Suppl 1:S9-S24).

In particular, Here below is provided the algorithm to compute each domain score:

- Effectiveness = [(item1 + item2 + item3) 3]/18\*100 = [(TSQM9\_1+TSQM9\_2+TSQM9\_3) 3]/18\*100
- Convenience = [(item4 + item5 + item6) 3]/18\*100 = [(TSQM9\_4+TSQM9\_5+TSQM9\_6) 3]/18\*100
- Global satisfaction = [(item7 + item8 + item9) 3]/14\*100 = [(TSQM9 7+TSQM9 8+TSQM9 9) 3]/14\*100

Each domain score can be calculated only if all the three items considered in the calculation of that score are not missing. Missing values will not be replaced.

The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain. Changes in the TSQM-9 subscale scores at each follow-up visit from enrollment will be calculated, for each patient, as the following difference: (subscales score at 6/12 months - subscale score at enrollment), if both scores are available.

#### MMAS-4 score

The Morisky medication Adherence Scale 4 items (MMAS-4) is a self-reported, medication-taking behavior scale and consists of four questions about the way patients might experience drug errors or omissions. Each item [F13\_MMAS\_4\_MMAS\_4\_1 - MMAS\_4\_4] has a scoring scheme of "Yes" = 0 and "No" = 1. Items are summed to give a non-adherence score ranging from 0 to 4; a higher score means better adherence to therapy (Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74).

The score can be calculated if at least 3 out of 4 of the items are completed. If only one item is omitted, the value for the missing item is the group median of this item that has been completed by all eligible participants. This median value will be imputed for all eligible cases who did not answer this item.

Changes in the MMAS-4 score at each follow-up visit from enrollment will be calculated, for each patient, as the following difference: (score at 6/12 months - score at enrollment), if both scores are available.

## COPD pharmacological treatments (classes) ongoing at enrollment

All COPD pharmacological treatments having "End date of therapy" [F20\_COPD\_PHARMACOLOGICAL\_THERAPY. END\_DATE\_THER] > "Date of enrollment visit" [\_PatientInfo.Date\_enrollment]) OR ("End date of therapy" missing and "Ongoing at the end of observation?" [F20\_COPD\_PHARMACOLOGICAL\_THERAPY. ONGOING\_THER] = "Yes"). Drug names will be coded by CDM and grouped according to the following categories:

- LAMA alone
- LABA alone

- ICS alone
- LABA + LAMA (Fixed dose combination or not)
- LABA + ICS (Fixed dose combination or not)
- LABA + LAMA + ICS
- SABA or SAMA on demand
- Other: pharmacological therapies for COPD not included in the previous classes.

Categories above are not mutally exclusive: a patient could be classified in more than one cathegory (i.e if a patient is receveing LAMA and SABA on demand, will be classified both in the "LAMA alone" and in the "SABA or SAMA on demand" classes). Only therapies for COPD will be considered (i.e. those records with field Therapy for [F20\_COPD PHARMACOLOGICAL THERAPY\_FOR] = "COPD"), while therapies for COPD exacerbations or for COPD-related adverse events will not be considered nor classified.

## COPD pharmacological treatments (classes) ongoing at 6- and 12-month follow-up visit

At each follow-up visit, all COPD treatments classes (see algorithm above) having

- ("Start date of therapy" [F20\_COPD PHARMACOLOGICAL THERAPY. START\_DATE\_THER] not missing AND < "Date of follow up visit" [F19\_PATIENT\_DISPOSITION. PD\_2]) AND</li>
- "End date of therapy" [F20\_COPD PHARMACOLOGICAL THERAPY. END\_DATE\_THER] not missing AND > "Date of follow up visit" [F19\_PATIENT\_DISPOSITION. PD\_2]) OR ("End date of therapy" missing AND "Ongoing at the end of observation?" [F20\_COPD PHARMACOLOGICAL THERAPY.ONGOING\_THER] = "Yes").

Drug names will be coded by CDM and grouped according to the categories specified above.

Only therapies for COPD will be considered (i.e. those records with field Therapy for [F20\_COPD PHARMACOLOGICAL THERAPY\_FOR] = "COPD"), while therapies for COPD exacerbations or for COPD-related adverse events will not be considered.

## COPD pharmacological treatments: fixed and non-fixed therapy

Patients with fixed COPD pharmacological treatments are those having at least one record of the COPD PHARMACOLOGICAL THERAPY form with "Is it a fixed dose combination?" [F20\_COPD PHARMACOLOGICAL THERAPY.DOSE\_2] = "Yes" for therapies ongoing at enrollment (see above).

Patients with non-fixed COPD pharmacological treatments are those having at least one record of the COPD PHARMACOLOGICAL THERAPY form with "Is it a fixed dose combination?" [F20\_COPD PHARMACOLOGICAL THERAPY.DOSE\_2] = "No" for therapies ongoing at enrollment (see above).

Patients who satisfy both conditions will be defined as **patients receiving both COPD pharmacological fixed and non-fixed therapy** at enrollment.

Data manager will check the congruence between the field "Drug" [F20\_COPD PHARMACOLOGICAL THERAPY.DRUG] and the question "Is it a fixed dose combination?": if any fixed dose drug will be entered in the field "Drug" and the question "Is it a fixed dose combination?" = "No" a query will be sent to the investigator. The vice-versa will be checked as well.

Only therapies for COPD will be considered, while therapies for COPD exacerbations or for COPD-related adverse events will not be considered.

## COPD pharmacological treatments: patients switching and not switching treatments

Considering only COPD pharmacological treatments (i.e. those records with field "Therapy for" [F20\_COPD PHARMACOLOGICAL THERAPY. THERAPY\_FOR] = "COPD") ongoing at enrollment or started after enrollment (i.e. with "Ongoing at the end of observation?" [F20\_COPD PHARMACOLOGICAL THERAPY. ONGOING\_THER] = "Yes" OR with "Start date of therapy" [F20\_COPD PHARMACOLOGICAL THERAPY. START\_DATE\_THER] > "Enrollment date"), patients who switched treatment during the observation period\* will be those with more than one record with the above-mentioned characteristics in the COPD PHARMACOLOGICAL THERAPY log form, excluding therapies started the very same day according to Start date of therapy. In particular, patients switching treatment are those with at least one change in the drug/frequency/route/formulation/device of administration after enrollment (also adding / stopping a COPD treatment is a switch).

\*switches occurred before enrollment will not be considered.

### Number of therapies administered for COPD, COPD-related adverse events and COPD exacerbations

The number of therapies administered for COPD per patient during observation period will be calculated as the sum of records of the COPD PHARMACOLOGICAL THERAPY log form considering only pharmacological treatments for COPD (i.e. those records with field "Therapy for" [F20\_COPD PHARMACOLOGICAL THERAPY. THERAPY\_FOR] = "COPD") ongoing at enrollment or started after enrollment (i.e. with "Ongoing at the end of observation?" [F20\_COPD PHARMACOLOGICAL THERAPY. ONGOING\_THER] = "Yes" OR with "Start date of therapy" [F20\_COPD PHARMACOLOGICAL THERAPY. START DATE THER] > "Enrollment date").

Similarly, the number of therapies administered for COPD-related adverse events and COPD exacerbations per patient during observation period will be calculated as the sum of records of the COPD PHARMACOLOGICAL THERAPY log form considering only pharmacological treatments for COPD-related adverse events and COPD exacerbations (i.e. those records with field "Therapy for" [F20\_COPD PHARMACOLOGICAL THERAPY. THERAPY\_FOR] = "COPD-related adverse event" OR "COPD exacerbation") ongoing at enrollment or started after enrollment (i.e. with "Ongoing at the end of observation?" [F20\_COPD PHARMACOLOGICAL THERAPY. ONGOING\_THER] = "Yes" OR with "Start date of therapy" [F20\_COPD PHARMACOLOGICAL THERAPY. START\_DATE\_THER] > "Enrollment date").

## **Exacerbations during the observation period**

Exacerbation is defined as "an increase or new onset of more than 1 symptom (cough, sputum, wheezing, dyspnoea or chest tightness) with at least 1 symptom lasting at least 3 days and leading to patient's attending physician to initiate treatment with systemic steroids and/or antibiotics (moderate exacerbation) or hospital admission (severe exacerbation)".

Patients with at least one exacerbation during observation period are those with "Did any exacerbation occur since the previous visit?" [F08\_EXACERBATIONS.EX\_Exacerbation\_YN] = "Yes", considering the 6- and 12-month follow-up visits and the End of observation visit.

The total number of exacerbations occurred during observation period per patient will be computed as the sum of the number of the matrix rows filled in the following fields: [F08\_EXACERBATIONS.Ex\_exacer\_1-10\_Ons\_date], considering the 6- and 12-month follow-up visits and the End of observation visit.

Hospitalizations for COPD, COPD exacerbations or COPD related adverse events during observation period. The total number of hospitalizations not in ICU for each patient will be the number of records in the matrix with "Patient admitted to intensive care unit?" [F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_ICU\_YN - RES\_Hosp\_matrix\_10\_\_ICU\_YN] = "No", considering the visit form HEALTHCARE RESOURCE CONSUMPTION at the 6- and 12-month follow-up visits and the End of observation visit.

The total number of hospitalizations in ICU for each patient will be the number of records in the matrix with "Patient admitted to intensive care unit?" [F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_ICU\_YN - RES\_Hosp\_matrix\_10\_\_ICU\_YN] = "Yes", considering the visit form HEALTHCARE RESOURCE CONSUMPTION at the 6- and 12-month follow-up visits and the End of observation visit.

The total number of days of hospitalization not in ICU for each patient will be the sum of the fields "Overall duration of admission (days)" [F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_Adm - RES\_Hosp\_matrix\_10\_\_Adm], considering only the records referred to hospitalizations not in ICU (see above) at the 6- and 12-month follow-up visits and the End of observation visit.

The total number of days of hospitalization in ICU for each patient will be the sum of the fields "Overall duration of admission (days)" [F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_Adm - RES\_Hosp\_matrix\_10\_\_Adm], considering only the records referred to hospitalizations in ICU (see above) at the 6- and 12-month follow-up visits and the End of observation visit.

ER accesses for COPD, COPD exacerbations or COPD related adverse events during observation period

The total number of ER accesses for each patient will be the sum of the fields "N° ER accesses" [F10\_RESOURCE\_CONS. RES\_ER\_matrix\_1\_\_n\_acc - RES\_ER\_matrix\_12\_\_n\_acc] considering the 6- and 12-month follow-up visits and the End of observation visit.

Specialist outpatient visits for COPD, COPD exacerbations or COPD related adverse events during observation period Patients with at least one specialist outpatient visit will be those with "Did the patient have any specialist outpatient visit for COPD, COPD exacerbations or COPD-related adverse events since the previous visit?" [F10\_RESOURCE\_CONS. RES\_OUTP\_YN] = "Yes" at 6-month follow-up visit OR at 12-month follow-up visits OR at End of observation visit.

The total number of specialist outpatient visits per patient during observation period will be computed as the sum of the field "Nr Visits" [F10\_RESOURCE\_CONS. RES\_Nr\_Visits], considering the 6- and 12-month follow-up visits and the End of observation visit.

General practitioner visits for COPD, COPD exacerbations or COPD related adverse events during observation period. The total number of general practitioner visits per patient during observation period will be computed as the sum of the field "N° of office visits (...)" [F10\_RESOURCE\_CONS. RES\_GP\_Visit\_YN\_Num], considering the 6- and 12-month follow-up visits and the End of observation visit.

Laboratory test for COPD, COPD exacerbations or COPD related adverse events during observation period. The total number of laboratory test per patient during observation period will be computed as the sum of the fields "N" of tests" [F10\_RESOURCE\_CONS. RES\_Lab\_matrix\_1\_num - RES\_Lab\_matrix\_20\_num] for each row of the matrix LABORATORY TESTS/EXAMINATIONS, considering the 6- and 12-month follow-up visits and the End of observation visit.

## Patients with oxygen therapy during the observational period

They will be defined as patients with at least one record in the OXYGEN THERAPY log form with ("Start date of therapy" [F21\_OXYGEN\_THERAPY. SART\_DATE\_NF] >= "Date of enrollment visit" [\_PatientInfo.Date\_enrollment] OR "Ongoing at the end of observation?" [F21\_OXYGEN\_THERAPY ONGOING\_NF\_THER] = "Yes").

## Patients with adverse events, serious adverse events, and adverse drug reactions

Patients with at least one adverse event (AE) will be those with at least one record in the AEs and ADRs log form with "AE brief description (in English)" [F22\_AES\_AND\_ADRS. AE\_DSCRPT] not missing.

**Patients with at least one serious adverse event (SAE)** will be those with at least one record in the AEs and ADRs log form with "AE brief description (in English)" not missing AND "Is it a serious AE?" [F22\_AES\_AND\_ADRS. AE\_1] = "Yes"

Patients with at least one adverse drug reaction (ADR) to one of the products marketed by Boheringer Ingelheim (namely: Spiriva Handihaler, Spiriva Respimat, Striverdi Respimat, Spiolto Respimat, Oxivent, Dosberotec, Duovent) will be those with at least one record in the AEs and ADRs log form with "AE brief description (in English)" not missing AND "Is there a reasonable causal relationship with one of the products marketed by Boheringer Ingelheim\*?" [F22 AES AND ADRS. AE 2] ="Yes".

#### 4 CONTENTS

The analyses will be performed on the Analysis set specified for each table.

Missing data will not be imputed and so patients with missing data will be excluded from the analyses of that variable(s). If the investigator is unable to collect the requested information the data will be "NK" (Not Known) or "NA" (Not Available), if the investigator did not record the information the data will be "Not Recorded".

## 4.1 Patient disposition

## Table 1. Enrolled and evaluable patients

The table will provide absolute and relative frequencies of:

- patients enrolled in the SAT study
- patients evaluable for safety analysis (Safety set) (as described in par. 2.4)
- patients evaluable at enrollment (Full analysis set) (as described in par. 2.1)
- patients evaluable at enrollment and at 6 month follow-up visit (as described in par. 2.2)
- patients evaluable at enrollment and at 12 month follow-up visit (as described in par. 2.3)

The percentages will be computed over the total number of enrolled patients.

### Table 2. Reasons for non-eligibility to analyses

The table will describe the reasons for patient non-eligibility.

Absolute and relative frequency distribution will be performed; the percentages will be computed out of the total number of enrolled patients.

### Table 3. Premature study termination

The table will describe the distribution of patients withdrawn from the study ("Did the patient complete the study?" [F18\_STUDY\_COMPLETION.SC\_1] = "No"); moreover, absolute and relative frequency of reasons for premature study termination ("Cause of drop out" [F18\_STUDY\_COMPLETION.SC\_2]) will be provided.

Percentages will be computed out of the total number of enrolled patients.

The distribution of patients withdrawn for other reasons will be also reported in a separate table ("If other cause, specify:" ≠ missing [F18\_STUDY\_COMPLETION.SC\_3]), if other reason frequency is >20%.

## 4.2 Demographics and baseline characteristics

## Table 4. Socio-demographic characteristics at enrollment

The table will provide:

- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' Age at enrollment
   ([ PatientInfo.Age])
- Patient distribution by Gender ([\_PatientInfo.Gender])
- Patient distribution by Race ([F02\_SOCIO\_DEMOGRAPHICS.SD\_Race])
- Patient distribution by Highest education level at baseline ([F02\_SOCIO\_DEMOGRAPHICS. SD\_Education])
- Patient distribution by Employment status at baseline ([F02\_SOCIO\_DEMOGRAPHICS. SD\_Employment])
- Patient distribution by Housing situation at baseline ([F02 SOCIO DEMOGRAPHICS.SD Housing])
- Patient distribution by Marital status at baseline ([F02 SOCIO DEMOGRAPHICS. SD Marital status])

Statistics will be computed out of the total number of FAS patients.

#### Table 5. Smoke habilts at enrollment

The table will provide:

- Patient distribution by Smoking status ([F03 LIFE HABITS.RF Smoking])
- Patient distribution by Kind of tobacco ([F03\_LIFE\_HABITS.RF\_Kind\_Tobacco])
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of the Estimated amount of tobacco consumed on average (pack/year) ([F03\_LIFE\_HABITS.RF\_Estimated\_amount\_Num])
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of Smoking duration in years (see 'Computed variables' chapter).

Percentages of smoking status will be computed out of the total number of FAS patients; for Kind of tobacco, Estimated amount of tobacco consumed on average, and Smoking duration, statistics will be computed over the total number of current / former smokers in the FAS.

#### Table 6. COPD medical history at enrollment

The table will provide:

- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of COPD duration at enrollment in years (see 'Computed variables' chapter)
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of age at COPD diagnosis (see 'Computed variables' chapter)
- Frequency distribution of Number of exacerbations in the last year at enrollment (in classes)
   ([F04 COPD\_MEDICAL\_HISTORY.MH\_nr\_exacerbations\_num])
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of Number of exacerbations in the last year at enrollment ([F04\_COPD\_MEDICAL\_HISTORY.MH\_nr\_exacerbations\_num])

Descriptives will be computed out of the total number of FAS patients.

#### Table 7. Comorbidities at enrollment

The table will provide the patient distribution by ongoing Comorbidity(ies) at enrollment (

([F06\_COMORBIDITIES.COM\_Comorbidities]). A patient could have more than one comorbidity.

Moreover, the patient distribution by Other comorbidities\* will be provided.

Percentages will be computed out of the total number of FAS patients .

## Table 8. Vital signs at enrollment

The table will provide:

- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' Weight at enrollment
   [F05 PHYSICAL EXAMINATION.PE Weight Num]
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' Height at enrollment [F05\_PHYSICAL\_EXAMINATION.PE\_Height\_Num]
- Patient distribution by BMI classes (see 'Computed variables' chapter)
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of BMI at enrollment [F05 PHYSICAL EXAMINATION. PE BMI]

Descriptives will be computed out of the total number of FAS patients.

## Table 9. Respiratory Functions at enrollment

The table will provide:

- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of FEV1 (L) at enrollment [F07 FUNCTIONAL ASSESSMENT.FA FEV1]
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of FEV1 of the predicted (%) at enrollment [F07 FUNCTIONAL ASSESSMENT.FA FEV1 predicted]
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of FVC (L) at enrollment [F07 FUNCTIONAL ASSESSMENT. FA FVC]
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of FEV1/FVC (%) at enrollment [F07\_FUNCTIONAL\_ASSESSMENT.FA\_FEV1\_FVC]
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of Residual Volume
   (L) at enrollment (F07 FUNCTIONAL ASSESSMENT.FA RV Num)
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of Inspiratory capacity (L) at enrollment [F07 FUNCTIONAL ASSESSMENT.FA VCIN Num]
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of Total lung capacity (L) at enrollment [F07\_FUNCTIONAL\_ASSESSMENT.FA\_TLC\_Num]
- Main descriptive statistics (mean, median, standard deviation, quartiles, min, max) of patients' values of DLCO at enrollment [F07\_FUNCTIONAL\_ASSESSMENT.FA\_DLCO\_Num], along with the respective DLCO unit [F07\_FUNCTIONAL\_ASSESSMENT.FA\_DLCO\_unit].

Descriptives will be computed out of the total number of FAS patients.

During data analysis, the Biostatistician will evaluate to perform the analyses described above also considering the evaluable patients at 6 months and/or at 12 months, depending on the number of patients of these analysis sets (in case the number of patients for these two analysis sets is relevantly different from the number of FAS patients), in order to understand if a selection bias is present.

## 4.3 Patients' satisfaction for medical treatment (TSQM-9) (primary objective)

## Table 10. Patients' satisfaction for medical treatment (TSQM-9 items) at each study visit

The table will provide absolute and relative frequency of patients' answers to TSQM-9 items (see Appendix 8.3) at each study visit.

Percentages will be calculated over the number of patients respectively evaluable at the time point considered, namely at enrollment (i.e. FAS patients), at 6 months (i.e. evaluable patients at 6 months) and at 12 months (i.e. evaluable patients at 12 months).

### Table 11. Patients' satisfaction for medical treatment (TSQM-9 subscales) at each study visit

The table will provide the descriptive statistics (mean, median, standard deviation, quartiles, min, max) of the TSQM-9 subscales scores (as defined in "Computed variables" chapter) at each study visit.

Changes from enrollment in TSQM-9 subscales scores (see 'Computed variables' chapter) will be also summarized by visit. 95% confidence intervals limits of the mean will be provided for each estimate (i.e. TSQM-9 subscales scores and changes). Descriptives will be calculated over the number of patients respectively evaluable at the time point considered, namely at enrollment (i.e. FAS patients), at 6 months (i.e. evaluable patients at 6 months) and at 12 months (i.e. evaluable patients at 12 months)

## 4.4 Patients' disease perception (B-IPQ) (secondary objective #1)

## Table 12. Patients' disease perception (B-IPQ) at each study visit

The table will provide the descriptive statistics (mean, median, standard deviation, quartiles, min, max) of B-IPQ questionnaire total score (as defined in "Computed variables" chapter) at each study visit.

Changes from enrollment in B-IPQ total score (see 'Computed variables' chapter) will be also summarized by visit.

95% confidence intervals limits of the mean will be provided for each estimate.

Descriptives will be calculated over the number of patients respectively evaluable at the time point considered, namely at enrollment (i.e. FAS patients), at 6 months (i.e. evaluable patients at 6 months) and at 12 months (i.e. evaluable patients at 12 months).

## 4.5 Patients' adherence to COPD treatment (MMAS-4) (secondary objective #1)

#### Table 13. Patients' adherence to COPD treatment (MMAS-4) at each study visit

The table will provide patient distribution by MMAS-4 answers to items #1-4 (Yes/No) at each study visit.

95% confidence intervals limits will be provided for each proportion. Moreover descriptive statistics (mean, median, standard deviation, quartiles, min, max) of MMAS-4 questionnaire total score (as defined in "Computed variables" chapter) at each study visit.

Changes from enrollment in MMAS-4 total score (see 'Computed variables' chapter) will be also summarized by visit.

Descriptives will be calculated over the number of patients respectively evaluable at the time point considered, namely at enrollment (i.e. FAS patients), at 6 months (i.e. evaluable patients at 6 months) and at 12 months (i.e. evaluable patients at 12 months).

(Missing values will be replaced according scoring algorithm as defined in "Computed variables" chapter, maximum one missing value is accepted).

## 4.6 Patients' health status (CAT) (secondary objective #1)

## Table 14. Patients' health status (CAT) at each study visit

The table will provide patient distribution by CAT questionnaire total score (as defined in "Computed variables" chapter, considering the following categories: < 10 / 10 - 20 / 21 - 30 / > 30) at each study visit.

The table will also provide the descriptive statistics (mean, median, standard deviation, quartiles, min, max) of CAT questionnaire total score (as defined in "Computed variables" chapter) at each study visit. Changes from enrollment in CAT total score (see 'Computed variables' chapter) will be also summarized by visit. 95% confidence intervals limits of the mean will be provided for each estimate.

Descriptives will be calculated over the number of patients respectively evaluable at the time point considered, namely at enrollment (i.e. FAS patients), at 6 months (i.e. evaluable patients at 6 months) and at 12 months (i.e. evaluable patients at 12 months).

(Missing values will be replaced according scoring algorithm as defined in "Computed variables" chapter, maximum two missing values are accepted).

## 4.7 Patients' dyspnea (mMRC) (secondary objective #1)

## Table 15. Patients' dyspnea (mMRC) at each study visit

Absolute and relative frequency of the mMRC grade at each study visit **[F15\_MMRC.MMRC]** (see Appendix 8.2); percentages will be calculated over the number of patients respectively evaluable at the time point considered, namely at enrollment (i.e. FAS patients), at 6 months (i.e. evaluable patients at 6 months) and at 12 months (i.e. evaluable patients at 12 months). 95% confidence intervals limits will be provided for each proportion.

#### 4.8 Patients' COPD awareness

## Table 16. Patients' COPD awareness (Awareness structured interview) each study visit

The table will provide:

- absolute and relative frequencies of patients' answers to each the COPD awareness questionnaire item
   [F12\_AWARENESS\_01 AWARENESS\_27] at each study visit;
- the descriptive statistics (mean, median, standard deviation, quartiles, min, max) of the COPD awareness questionnaire composite scores (see 'Computed variables' chapter) at each study visit.

Changes from enrollment in the COPD awareness composite scores (see 'Computed variables' chapter) will be also summarized by visit.

95% confidence intervals limits of the mean will be provided for each estimate.

Descriptives will be calculated over the number of patients respectively evaluable at the time point considered, namely at enrollment (i.e. FAS patients), at 6 months (i.e. evaluable patients at 6 months) and at 12 months (i.e. evaluable patients at 12 months).

# 4.9 Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period (secondary objective #2)

The purpose of this secondary analysis is not to obtain a predictive model, but to investigate the relationship among pre-defined variables and outcomes that are of clinical interest. In fact, the intent of this analysis is mainly exploratory and not confirmatory of any a priori hypotheses (consistently with the Study Protocol indications).

Among independent variables in the model, the PROs used in the study are symptomatic tools routinely used in clinical practice to evaluated disease activity and severity (i.e. mMRC and CAT) as per the patient's perspective. Patients' treatment satisfaction could also depend on their clinical status (that would be measured through the mMRC or the CAT) and on their adherence to treatment (MMAS-4 score). This is the reason why the PROs measures are taken into account in exploring the relationship between patient's treatment satisfaction and clinical status.

Contrary to what is stated in paragraph 9.7 of the Study Protocol, the Sponsor on the 12/09/2017 decided not to include the covariates post-baseline in this analysis: therefore, only data collected at enrollment visit will be considered in the mixed models for repeated measures described below, with the exception of the dependent variables (i.e. TSQM-9 scores, that will be considered at each timepoint).

## Table 17. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period (Repeated measures regression models) – Effectiveness domain

A regression model will be estimated; the dependent variable will be the effectiveness domain score of TSQM-9 and the independent ones will be the following:

- age and gender at enrollment;
- number of exacerbations at enrollment;
- relevant spirometry parameters at enrollment (a selection of the following parameter will be done, based on data availability: FEV1, FVC, FEV1 % of the predicted, RV, TLC, DLCO);
- patient's disease severity in terms of level of dyspnea (mMRC score) or CAT total score (depending on data availability) at enrollment (since they are expected to be intercorrelated measures, as reported by 2017 GOLD guidelines, only one of such measures will be considered in the model);
- MMAS-4 score at enrollment.

Center will be included as random effect and study visit (visit1/enrollment, visit2/6months, and visit3/12months) as timepoint. During data elaboration, the Biostatistician will assess the intercorrelation between the proposed variables, in order to evaluate the opportunity to exclude some of the listed independent variables that are highly associated to each other; in case of important lack of data for certain parameters, such parameters may be excluded as well from the final model.

Because measures referred to the dependent variable will be collected at each study visit, a mixed model for repeated measures will be estimated; moreover, interaction terms between independent variables will be evaluated and, if not significant, they will not be included in the final model. The optimal covariance structure will be evaluated during analysis (preferably "first-order autoregressive correlation" or "unstructured" options). A stepwise selection method will be evaluated during the analysis in order to identify the variables to be included in the final model.

The patients switching treatment during observation period will not be excluded from analysis. The patients stopping treatment during study will be censored at last available visit.

The analysis will be performed considering only evaluable patients at 12 months.

## Table 18. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period (Repeated measures regression models) – Convenience domain

See previous model characteristics: in this analysis, the dependent variable will be the convenience domain score of TSQM-9.

## Table 19. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period (Repeated measures regression models) – Global satisfaction domain

See previous model characteristics: in this analysis, the dependent variable will be the global satisfaction domain score of TSQM-9.

## 4.10 Healthcare resource utilization (secondary objective #3)

## Table 20. Hospitalizations not in ICU during observation period: patients' distribution

The table will provide:

- distribution of patients by number of hospitalization not in ICU per patient during observation period (see 'Computed variables' chapter);
- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of number of hospitalization not in ICU during observation period per patient (see 'Computed variables' chapter);
- distribution of patients by "Type of admission" ([F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_Inw RES\_Hosp\_matrix\_10\_\_Inw]), considering only hospitalization not in ICU according to the field [RES\_Hosp\_matrix\_x\_ICU\_YN];
- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of total number of days of hospitalization not in ICU per patient (see 'Computed variables' chapter);
- distribution of patients by reasons for hospitalization not in ICU (i.e. "Hospitalization for" [F10\_RESOURCE\_CONS.
   RES\_Hosp\_matrix\_1\_hos\_for RES\_Hosp\_matrix\_10\_hos\_for]).

Descriptives and percentages will be computed out of the total number of FAS patients.

## Table 21. Hospitalizations not in ICU during observation period: details

The table will provide:

- distribution of hospitalizations not in ICU by "Type of admission" ([F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_Inw RES\_Hosp\_matrix\_10\_\_Inw]), considering only hospitalization not in ICU according to the field [RES\_Hosp\_matrix\_x\_ICU\_YN];
- distribution of hospitalizations not in ICU by reasons for hospitalization (i.e. "Hospitalization for" [F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_hos\_for RES\_Hosp\_matrix\_10\_\_hos\_for]).

Statistics will be computed out of the total number of hospitalizations not in ICU during observation period in FAS patients.

## Table 22. Hospitalizations in ICU during observation period: patients' distribution

The table will provide:

- distribution of patients by number of hospitalization in ICU during observation period (see 'Computed variables' chapter);
- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of number of hospitalization in ICU during observation period per patient (see 'Computed variables' chapter);
- distribution of patients by "Type of admission" ([F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_Inw RES\_Hosp\_matrix\_10\_\_Inw]), considering only hospitalization in ICU according to the field [RES Hosp matrix x ICU YN];
- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of total number of days of hospitalization in ICU (see 'Computed variables' chapter);
- distribution of patients by reasons for hospitalization in ICU (i.e. "Hospitalization for" [F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_hos\_for RES\_Hosp\_matrix\_10\_\_hos\_for]).

Descriptives and percentages will be computed out of the total number of FAS patients.

## Table 23. Hospitalizations in ICU during observation period: details

The table will provide:

- distribution of hospitalizations in ICU by "Type of admission" ([F10\_RESOURCE\_CONS. RES\_Hosp\_matrix\_1\_\_Inw RES\_Hosp\_matrix\_10\_\_Inw]), considering only hospitalization in ICU according to the field [RES\_Hosp\_matrix\_x\_ICU\_YN];
- distribution of hospitalizations in ICU by reasons for hospitalization (i.e. "Hospitalization for"
   [F10 RESOURCE CONS. RES Hosp matrix 1 hos for RES Hosp matrix 10 hos for]).

Statistics will be computed out of the total number of hospitalizations in ICU during observation period in FAS patients.

## Table 24. Emergency room accesses: patients' distribution

The table will provide:

distribution of patients by number of ER accesses during observation period per patient (see 'Computed variables' chapter);

- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of number of ER accesses during observation period per patient (see 'Computed variables' chapter);
- distribution of patients by reasons of ER admission (i.e. "Admission for" [F10\_RESOURCE\_CONS.
   RES ER matrix 1 adm for RES ER matrix 12 adm for]).

Descriptives and percentages will be computed out of the total number of FAS patients.

## Table 25. Emergency room accesses: details

The table will provide:

distribution of reasons of ER accesses during observation period (i.e. "Admission for" [F10\_RESOURCE\_CONS.
 RES\_ER\_matrix\_1\_\_adm\_for - RES\_ER\_matrix\_12\_\_adm\_for]).

Statistics computed over the total number of ER accesses during observation period in FAS patients.

## Table 26. Specialist outpatient visits: patients' distribution

The table will provide:

- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of the total number of specialist outpatient visits per patient during observation period (see 'Computed variables' chapter);
- distribution of patients by number of specialist outpatient visits per patient during observation period (see 'Computed variables' chapter);
- distribution of patients by type of specialist outpatient visits performed during observation period (i.e. "Specialist "[F10 RESOURCE CONS. Specialist]);
- distribution of patients by reasons of specialist outpatient visit (i.e. "Visit for" [F10\_RESOURCE\_CONS. RES\_Visit\_for]).

Descriptives and percentages will be computed out of the total number of FAS patients.

## Table 27. General practitioner visits: patients' distribution

The table will provide:

- distribution of patients by total number of general practitioner visits per patient during observation period (see 'Computed variables' chapter);
- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of the total number of general practitioner visits per patient during observation period (see 'Computed variables' chapter).

Descriptives and percentages will be computed out of the total number of FAS patients.

## Table 28. Laboratory tests: patients' distribution

The table will provide:

- distribution of patients by total number of laboratory test per patient during observation period (see 'Computed variables' chapter);
- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of total number of laboratory test per patient during observation period (see 'Computed variables' chapter);
- distribution of patients by type of test/examination during observation period (i.e. "Test/examination" [F10\_RESOURCE\_CONS. RES\_Lab\_matrix\_1\_Test RES\_Lab\_matrix\_20\_Test]);
- distribution of patients by reasons of test/examination (i.e. "Test/examination for" [F10\_RESOURCE\_CONS.
   RES Lab matrix 1 for RES Lab matrix 20 for]).

Descriptives and percentages will be computed out of the total number of FAS patients.

#### Table 29. Laboratory tests: details

The table will provide:

- frequency of each type of test/examination during observation period (listed in field "Test/examination" [F10\_RESOURCE\_CONS. RES\_Lab\_matrix\_1\_Test RES\_Lab\_matrix\_10\_Test] and according to the number of tests recorded in field "N° of tests" [F10\_RESOURCE\_CONS. RES\_Lab\_matrix\_1\_num RES\_Lab\_matrix\_20\_num]),
- distribution of reasons of test/examination (i.e. "Test/examination for" [F10\_RESOURCE\_CONS. RES\_Lab\_matrix\_1\_for - RES\_Lab\_matrix\_20\_for]).

Statistics computed over the total number of Laboratory tests during observation period in FAS patients.

## Table 30. Oxygen therapy

The table will provide:

Absolute and relative frequency of Patients with oxygen therapy during the observational period (see 'Computed variables' chapter)

Percentages will be computed out of the total number of patients evaluable for the FAS.

## Table 31. List of oxygen therapies

List of the following variables:

- Patient ID
- "Date of enrollment visit" [ PatientInfo.Date enrollment]
- "Kind of therapy" [F21\_OXYGEN\_THERAPY.KIND\_OF\_THER]
- "Drug" [F21\_OXYGEN\_THERAPY.DRUG]
- "Flow (L/min)" [F21\_OXYGEN\_THERAPY.FLOW]
- "Hours per day" [F21\_OXYGEN\_THERAPY.HOURS]
- "Start date of therapy" [F21\_OXYGEN\_THERAPY.START\_DATE\_NF]
- "Ongoing" [F21\_OXYGEN\_THERAPY.ONGOING\_NF\_THER]
- "End date of therapy" [F21\_OXYGEN\_THERAPY.END\_DATE\_NF]
- "Therapy for" [F21 OXYGEN THERAPY.NF THER FOR]

Only patients evaluable for the FAS will be considered.

### Table 32. Patients receiving fixed/non-fixed dose therapies for COPD at enrollment

The table will provide:

- distribution of patients with COPD pharmacological fixed dose therapy at enrollment (see 'Computed variables' chapter);
- distribution of patients with COPD pharmacological non-fixed dose therapy at enrollment (see 'Computed variables' chapter);
- distribution of patients receiving both COPD pharmacological fixed and non-fixed therapy at enrollment (see 'Computed variables' chapter).

Percentages will be computed out of the total number of patients evaluable for the FAS.

## Table 33. COPD pharmacological treatments ongoing at enrollment

The table will provide:

• distribution of COPD pharmacological treatments (classes) ongoing at enrollment (see 'Computed variables' chapter). Percentages will be computed out of the total number of patients evaluable for the FAS.

#### Table 34. COPD pharmacological treatments ongoing at 6-month follow-up visit

The table will provide:

distribution of COPD pharmacological treatments (classes) ongoing at 6-month follow-up visit (see 'Computed variables' chapter)

Percentages will be computed out of the total number of patients evaluable for the FAS.

### Table 35. COPD pharmacological treatments ongoing at 12-month follow-up visit

The table will provide:

distribution of COPD pharmacological treatments (classes) ongoing at 12-month follow-up visit (see 'Computed variables' chapter)

Percentages will be computed out of the total number of patients evaluable for the FAS.

## Table 36. Medications for adverse events

The table will provide the distribution of patients according to the field "Therapy for the event" [F22\_AES\_AND\_ADRS. AE\_THERAPY] (i.e. patients who received medications for adverse events during the study).

Percentages will be computed out of the total number of patients evaluable for the FAS.

## 4.11 Correlation between patients' satisfaction and resource utilization (secondary objective #4)

## Table 37. Correlation between patients' satisfaction and resource utilization (including drugs)

A correlation index (Pearson or Spearman) will be computed between TSQM-9 subscales scores (as defined in "Computed variables" chapter) at 12 month follow-up visit and the number of hospitalizations per patient during observation period (as defined in "Computed variables" chapter); p-value will be provided as well.

A correlation index (Pearson or Spearman) will be computed between TSQM-9 subscales scores (as defined in "Computed variables" chapter) at 12 month follow-up visit and the number of ER accesses per patient during observation period (as defined in "Computed variables" chapter); p-value will be provided as well.

A correlation index (Pearson or Spearman) will be computed between TSQM-9 subscales scores (as defined in "Computed variables" chapter) at 12 month follow-up visit and the number of specialist visits per patient during observation period (as defined in "Computed variables" chapter); p-value will be provided as well.

A correlation index (Pearson or Spearman) will be computed between TSQM-9 subscales scores (as defined in "Computed variables" chapter) at 12 month follow-up visit and the number of general practitioner visits per patient during observation period (as defined in "Computed variables" chapter); p-value will be provided as well.

A correlation index (Pearson or Spearman) will be computed between TSQM-9 subscales scores (as defined in "Computed variables" chapter) at 12 month follow-up visit and the number of laboratory test per patient during observation period (as defined in "Computed variables" chapter); p-value will be provided as well.

A correlation index (Pearson or Spearman) will be computed between TSQM-9 subscales scores (as defined in "Computed variables" chapter) at 12 month follow-up visit and the number of therapies administered for COPD per patient during observation period (as defined in "Computed variables" chapter); p-value will be provided as well.

A correlation index (Pearson or Spearman) will be computed between TSQM-9 subscales scores (as defined in "Computed variables" chapter) at 12 month follow-up visit and the number of therapies administered for COPD-related adverse events and COPD exacerbations per patient during observation period (as defined in "Computed variables" chapter); p-value will be provided as well.

#### 4.12 Exacerbations

#### Table 38. Exacerbations: patients' distribution

This table will provide:

- the distribution of patients by number of exacerbations per patient during observation period (see 'Computed variables' chapter);
- descriptive statistics (mean, median, standard deviation, quartiles, min, max) of number of exacerbations per patient during observation period (see 'Computed variables' chapter);
- the distribution of patients by exacerbation severity [F08\_EXACERBATIONS. Ex\_Exacer\_1\_severity Ex\_Exacer\_10\_severity];
- the distribution of patients by changes in COPD therapy due to exacerbations (i.e. "Any new therapy or any change to an ongoing one required\*?" [F08\_EXACERBATIONS. Ex\_Exacer\_1\_change Ex\_Exacer\_10\_change]).

Percentages will be computed out of the total number of patients evaluable for the FAS.

#### Table 39. Exacerbations: details

This table will provide:

- the distribution of exacerbations by exacerbation severity [F08\_EXACERBATIONS. Ex\_Exacer\_1\_severity Ex Exacer 10 severity];
- the distribution of exacerbations by changes in COPD therapy due to exacerbations (i.e. "Any new therapy or any change to an ongoing one required\*?" [F08\_EXACERBATIONS. Ex\_Exacer\_1\_change Ex Exacer 10 change]).

Percentages will be computed out of the total number of exacerbations occurred during observation period in FAS patients.

## 4.13 Safety

### Table 40. Overall Summary of Adverse Events and Adverse Event Reactions

This table will provide:

- the absolute and relative frequency of patients with at least one adverse event (AE) (see 'Computed variables' chapter),
- the absolute and relative frequency of patients with at least one Serious Adverse Event (SAE) (see 'Computed variables' chapter), and
- the patients distribution by "Seriousness Category" [F22\_AES\_AND\_ADRS. AE\_SERIOUSNESS\_CAT], and
- the absolute and relative frequency of patients with at least one Adverse Drug Reaction (ADR) to one of the products marketed by Boheringer Ingelheim (namely: Spiriva Handihaler, Spiriva Respimat, Striverdi Respimat, Spiolto Respimat, Oxivent, Dosberotec, Duovent) (see 'Computed variables' chapter), and
- the patients distribution by "Product" [F22\_AES\_AND\_ADRS. AE\_BI\_Product]

over the total number of evaluable patients for the Safety set.

## Table 41. Patients' distribution by type of adverse event

This table will provide the patients distribution by type of adverse events (i.e. "AE brief description (in English)" [F22\_AES\_AND\_ADRS.AE\_DSCRPT].

Percentages will be computed over the total number of evaluable patients for the Safety set.

## Table 42. Distribution of type of adverse event: details

This table will provide the frequency of each type of adverse events (i.e. "AE brief description (in English)" [F22\_AES\_AND\_ADRS.AE\_DSCRPT].

Percentages will be computed over the total number of AEs occurred in the Safety set.

#### Table 43. List of adverse events

The list of all adverse events occurred in the Safety set will be reported. The following variables will be described:

- Patient ID
- "Date of enrollment visit" [\_PatientInfo.Date\_enrollment]
- "AE brief description (in English)" [F22\_AES\_AND\_ADRS.AE\_DSCRPT]
- "Date of onset" [F22 AES AND ADRS.AE ONSET]
- "Is it ongoing at the end of the study?" [F22\_AES\_AND\_ADRS.AE\_ONGOING]
- "End date" [F22\_AES\_AND\_ADRS.AE\_END\_DATE]
- "Is it a serious AE" [F22 AES AND ADRS.AE 1]
- "Seriousness category" [F22\_AES\_AND\_ADRS.AE\_SERIOUSNESS\_CAT]
- "Is there a reasonable causal relationship with one of the products marketed by BI?" [F22 AES AND ADRS.AE 2]
- "Product" [F22\_AES\_AND\_ADRS.AE\_BI\_PRODUCT]
- "Action taken with BI drug" [F22\_AES\_AND\_ADRS.AE\_ACTION]
- "Therapy for the event" [F22\_AES\_AND\_ADRS.AE\_THERAPY]
- "Outcome of the event" [F22\_AES\_AND\_ADRS.AE\_OUTCOME]

#### Table 44. Pregnancies: patients' distribution

This table will provide the patients distribution according to the field "Pregnancy" [F23\_PREGNANCY. PREGNANCY\_1] over the total number of evaluable patients for the Safety set.






















































#### 6 QUALITY CHECKS ON THE STATISTICAL REPORT

The statistical analysis of the SAT study will be managed by 3 main figures in the Biostatistician (BS), the Clinical Data Manager (CDM) and the Manager of Data Management and Statistics unit (R-DMS). In particular, in this context, CDM is the owner of data cleaning, database creation, management and lock, while BS is the owner of Statistical Analysis Plan and Statistical Report redaction.

BS and CDM of the SAT study have performed an annual training of at least 30 hours and an induction training concerning knowledge and skills required for the management of observational studies with a focus on their role. Furthermore they are coordinated by R-DMS who possesses qualifications necessary for job.

Moreover, regarding instruments, database management and data analysis will be performed using SAS Enterprise Guide v. 7.1 and SAS 9.4.

Actions to improve the quality of data are taken in different moments during the study and using various tools, as described in Standard Operating Procedures concerning data cleaning and statistical analysis.

Data validation (see Data Validation Plan) foresees both on-line (electronic CRF allows to verify data at the moment they are entered by means of automated edit checks, out of range controls, etc.) and off-line checks. Subsequently, quality control continues at the moment of the database lock when, as requested by procedure, the CDM can lock the database only if, among other conditions, BS and Sponsor approve the quality of data (i.e. In defining if the obtained quality of data is sufficient, the impact of possible missing/inconsistent data remained after all possible efforts to fix are done, will be based on the impact of these data on the primary and the secondary study objectives).

Finally, a quality control of the data analysis process focused on the detection of possible calculation errors or inconsistent data is performed. To observe the recommendation about the detection of priorities in order to make the process more efficient, the type of statistical report quality control is defined on the basis of the risk analysis conducted for the study.

The following quality controls will be performed on the statistical report of the SAT study.

- All the tables described in this document will be programmed and verified by a BS.
- R-DMS will perform an overall conceptual review of results, in order to evaluate their coherence and plausibility. Moreover, all the tables in this report will be independently reviewed to verify their consistency.
- Moreover, the following tables will be reprogrammed or independently verified (by another BS or CDM):
  - **Table 93. Enrolled and evaluable patients:** 100% of patients will be checked by a CDM or another BS in order to assess whether the evaluability variables are correctly computed according to the algorithm described in the SAP.
  - **Table 2. Reasons for non-eligibility to analyses:** 100% of patients will be checked by a CDM or another BS in order to assess whether the evaluability variables are correctly computed according to the algorithm described in the SAP.
  - **Table 3. Premature study termination:** 100% of patients will be checked by a CDM or another BS in order to verify the number of completed/discontinued patients and frequency of cause of drop-out.
  - Table 4. Socio-demographic characteristics at enrollment: Table output will be verified by another BS or CDM
  - **Table 5. Smoke habilts at enrollment:** Table output will be verified by another BS or CDM; moreover, smoking duration will be verified by CDM/another BS in order to assess if it is computed according to the algorithm described in the SAP
  - Table 6. COPD medical history at enrollment: Table output will be verified by another BS or CDM; moreover, COPD duration and age at COPD diagnosis will be verified by CDM/another BS in order to assess if it is computed according to the algorithm described in the SAP
  - Table 7. Comorbidities at enrollment: Table output will be verified by another BS or CDM
  - Table 8. Vital signs at enrollment: Table output will be verified by another BS or CDM
  - Table 11. Patients' satisfaction for medical treatment (TSQM-9 subscales) at each study visit: another BS/CDM will verify 100% of evaluable patients in order to assess that the TSQM-9 subscales scores are calculated according to the algorithm described in the SAP
  - **Table 12. Patients' disease perception (B-IPQ) at each study visit**: randomly chosen patients (50% of evaluable patients) will be checked by a CDM or another BS in order to assess whether B-IPQ total score is correctly computed according to the algorithm described in the SAP.
  - Table 13. Patients' adherence to COPD treatment (MMAS-4) at each study visit: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (50% of evaluable patients) will be checked by a CDM or another BS in order to assess whether MMAS-4 total score is correctly computed according to the algorithm described in the SAP.
  - **Table 14. Patients' health status (CAT) at each study visit:** randomly chosen patients (50% of evaluable patients) will be checked by a CDM or another BS in order to assess whether CAT total score is correctly computed according to the algorithm described in the SAP.
  - Table 16. Patients' COPD awareness (Awareness structured interview) each study visit: randomly chosen patients (50% of evaluable patients) will be checked by a CDM or another BS in order to assess whether COPD awareness questionnaire's composite scores are correctly computed according to the algorithm described in the SAP.
  - Table 19. Relation between treatment satisfaction and demographic/clinical parameters and PROs during 12 month observation period (Repeated measures regression models) Global satisfaction domain: another BS will verify the results obtained from the mixed model for repeated measures

- Table 20. Hospitalizations not in ICU during observation period: patients' distribution: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (20% of evaluable patients) will be checked by a CDM or another BS in order to assess whether Number of hospitalization not in ICU during observation period per patient and Number of days of hospitalization not in ICU per patient are correctly computed according to the algorithm described in the SAP
- Table 23. Hospitalizations in ICU during observation period: details: Table output will be verified by another BS or CDM
- Table 24. Emergency room accesses: patients' distribution: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (20% of evaluable patients) will be checked by a CDM or another BS in order to assess whether Number of ER accesses during observation period per patient is correctly computed according to the algorithm described in the SAP
- Table 26. Specialist outpatient visits: patients' distribution: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (20% of evaluable patients) will be checked by a CDM or another BS in order to assess whether Number of specialist outpatient visits per patient during observation period is correctly computed according to the algorithm described in the SAP
- Table 27. General practitioner visits: patients' distribution: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (20% of evaluable patients) will be checked by a CDM or another BS in order to assess whether Number of general practitioner visits per patient during observation period is correctly computed according to the algorithm described in the SAP
- **Table 28. Laboratory tests: patients' distribution**: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (20% of evaluable patients) will be checked by a CDM or another BS in order to assess whether Number of laboratory tests/examinations per patient during observation period is correctly computed according to the algorithm described in the SAP
- Table 30. Oxygen therapy: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (10% of evaluable patients) will be checked by a CDM or another BS in order to assess whether Patients with oxygen therapy during the observational period were correctly identified according to the algorithm described in the SAP
- **Table 31. List of oxygen therapies**: 3 patients will be verified with respect to DB content
- Table 32. Patients receiving fixed/non-fixed dose therapies for COPD ongoing at enrollment: randomly chosen patients (10% of evaluable patients) will be checked by a CDM or another BS in order to assess whether patients with COPD pharmacological fixed and/or non-fixed dose therapy ongoing at enrollment were correctly identified according to the algorithm described in the SAP
- **Table 33. COPD pharmacological treatments ongoing at enrollment:** randomly chosen patients (10 for each COPD pharmacological treatment cathegory) will be checked by a CDM or another BS in order to assess whether the patient was correctly classified according to the algorithm described in the SAP.
- Table 37. Correlation between patients' satisfaction and resource utilization (including drugs): another BS will verify the correlations coefficients and p-values
- **Table 38. Exacerbations: patients' distribution**: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (20% of evaluable patients) will be checked by a CDM or another BS in order to assess whether Number of exacerbations per patient during observation period is correctly computed according to the algorithm described in the SAP
- Table 40. Overall Summary of Adverse Events and Adverse Event Reactions: Table output will be verified by another BS or CDM; moreover, randomly chosen patients (10% of evaluable patients) will be checked by a CDM or another BS in order to assess whether patients with at least one AE/SAE/ADR were correctly identified according to the algorithm described in the SAP
- Table 43. List of adverse events: 3 patients will be verified with respect to DB content
- Table 45. Patients' satisfaction for medical treatment (TSQM-9 items) at each study visit Switchers vs non-switchers: randomly chosen patients (50% of evaluable patients) will be checked by a CDM or another BS in order to assess whether they were correctly classified as switchers/non-switchers.

# 7 REVISION HISTORY

| Table (N° and title) | SAP version and date | Change description | Applicant | Note |
|---|---|---|---|---|
| All applicable tables | Vers.1.0,<br>16/09/2016 | Analysis modified according to the changes agreed with Sponsor during the conference call held on the 27/09/2016 | BI | |
| All applicable tables | Vers.1.0,<br>16/09/2016 | General review of the document and proposed analyses | | |
| Whole document | Vers.1.1,<br>10/07/2017 | General review of the document | Bl Global | |
| Tables 4-6 | Vers. 1.2,<br>25/07/2017 | Descriptive analyses on non-evaluable patients removed | BI Global | |
| Tables 20-22 | Vers. 1.2,<br>25/07/2017 | Regression model characteristics further specified | BI Global, | |
| Whole document | Vers. 1.3,<br>15/09/2017 | General review of the document | Bl Global | |
| Table 14 | Vers. 1.4,<br>21/09/2017 | Analysis on CAT score categories added | Bl Global | |

#### 8 APPENDICES

### 8.1 COPD awareness questionnaire scoring system

The following table specifies the score that is to be given to the single answer options of each COPD awareness questionnaire's item.

| 90.0 | Stiormane's item. | Domain | Per nulla<br>d'accordo | Poco<br>d'accordo | Abbastanza<br>d'accordo | Molto<br>d'accordo |
|---|---|---|---|---|---|---|
| 1. | Dovrò assumere i farmaci inalatori per sempre | Knowledge of disease | 0 | 1 | 2 | 3 |
| 2. | Penso che la BPCO tenda a peggiorare con il passare del tempo | Knowledge of disease | 0 | 1 | 2 | 3 |
| 3. | I farmaci per la BPCO mi permettono di svolgere le normali attività quotidiane | - | 0 | 1 | 2 | 3 |
| 4. | I farmaci presi regolarmente permettono di muoversi con minor fatica | Awareness of treatment needs | 0 | 1 | 2 | 3 |
| 5. | Penso che la BPCO sia una malattia poco grave, infatti viene curata con farmaci per inalazione | Disease perception | 3 | 2 | 1 | 0 |
| 6. | Il fumo è la causa principale della BPCO | - | 0 | 1 | 2 | 3 |
| 7. | Faccio fatica ad accettare di avere la BPCO | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 8. | I farmaci somministrati per via inalatoria sono meno potenti delle pillole, compresse o altre medicine prese per bocca | Disease perception | 3 | 2 | 1 | 0 |
| 9. | I farmaci per la BPCO vanno presi regolarmente | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 10. | Preferisco ignorare i sintomi della BPCO | Disease perception | 3 | 2 | 1 | 0 |
| 11. | I farmaci inalatori possono essere sospesi quando i sintomi migliorano | - | 3 | 2 | 1 | 0 |
| 12. | La terapia regolare riduce i peggioramenti improvvisi | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 13. | E' normale, alla mia età, avere problemi respiratori | - | 3 | 2 | 1 | 0 |
| 14. | I farmaci assunti per via inalatoria consentono di migliorare la fatica a respirare | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 15. | Sono preoccupato per la mia BPCO | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 16. | Da quando ho la BPCO faccio fatica a sentirmi me stesso | - | 3 | 2 | 1 | 0 |
| 17. | La sospensione della terapia inalatoria aumenta i peggioramenti | - | 0 | 1 | 2 | 3 |
| 18. | La spirometria è un esame fondamentale per giungere alla diagnosi di BPCO | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 19. | Penso che la mia BPCO non guarirà mai | Knowledge of disease | 0 | 1 | 2 | 3 |
| 20. | Penso che la mia BPCO non guarirà mai perché non ci sono farmaci efficaci | Disease perception | 3 | 2 | 1 | 0 |
| 21. | Preferisco non pensare al fatto di avere la BPCO | Disease perception | 3 | 2 | 1 | 0 |
| 22. | L'idea di soffrire di BPCO mi fa arrabbiare | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 23. | I farmaci per la BPCO migliorano i sintomi | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 24. | Faccio fatica a convivere con i sintomi della BPCO | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 25. | Mi chiedo perché questa malattia sia capitata proprio a me | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 26. | La BPCO è una malattia cronica, cioè non guarisce | Knowledge of disease | 0 | 1 | 2 | 3 |
| 27. | Tutti i fumatori soffrono di BPCO | - | 3 | 2 | 1 | 0 |

Here below, the meaning of each question and answer option in English language (which is not an official, validated translation) is provided:

| | | Domain | I totally<br>disagree | l agree a<br>little | I somewhat agree | l totally<br>agree |
|---|---|---|---|---|---|---|
| 1. | I need to be treated with inhaled drugs forever | Knowledge of disease | 0 | 1 | 2 | 3 |
| 2. | I believe that COPD tends to worsen over time | Knowledge of disease | 0 | 1 | 2 | 3 |
| 3. | Treatments for COPD allow me to carry out normal daily activities | - | 0 | 1 | 2 | 3 |
| 4. | A regular administration of drugs allows me to move with less effort | Awareness of treatment needs | 0 | 1 | 2 | 3 |
| 5. | I think that COPD is a mild disease since it is treated with inhaled drugs | Disease perception | 3 | 2 | 1 | 0 |
| 6. | Smoke is the main cause of COPD | - | 0 | 1 | 2 | 3 |
| 7. | I cannot easily accept to have COPD | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 8. | Inhaled drugs are less effective than pills, tablets or other oral medications | Disease perception | 3 | 2 | 1 | 0 |
| 9. | Treatments for COPD must be taken regularly | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 10. | I prefer to ignore COPD symptoms | Disease perception | 3 | 2 | 1 | 0 |
| 11. | Inhaled drugs can be interrupted if symptoms improve | - | 3 | 2 | 1 | 0 |
| 12. | A regular therapy reduces the risk of sudden worsening | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 13. | It is common to have respiratory problems at my age | - | 3 | 2 | 1 | 0 |
| 14. | Inhaled drugs help improving the fatigue in breathing | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 15. | I am worried about my COPD | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 16. | I have been finding it hard to feel like myself since I suffer from COPD | - | 3 | 2 | 1 | 0 |
| 17. | Interrupting the inhaled therapy increases the risk of COPD worsening | - | 0 | 1 | 2 | 3 |
| 18. | Spirometry is a fundamental examination for the COPD diagnosis | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 19. | I will never heal from my COPD | Knowledge of disease | 0 | 1 | 2 | 3 |
| 20. | I think I will never heal from my COPD because there is lack of effective drugs | Disease perception | 3 | 2 | 1 | 0 |
| 21. | I prefer not to think about my COPD | Disease perception | 3 | 2 | 1 | 0 |
| 22. | I am angry because of my COPD | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 23. | Drugs for COPD improve my symptoms | Awareness of<br>treatment needs | 0 | 1 | 2 | 3 |
| 24. | I am having difficulty living with COPD symptoms | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 25. | I wonder why COPD happened to me | Acknowledgement of disease | 3 | 2 | 1 | 0 |
| 26. | COPD is a chronic disease and it is not possible to heal from it | Knowledge of disease | 0 | 1 | 2 | 3 |
| 27. | All smokers suffer from COPD | - | 3 | 2 | 1 | 0 |

#### 8.2 Modified Medical Research Council (mMRC) dyspnoea scale

- Italian version (used in the SAT study)

# Scala modificata del Medical Research Council (mMRC) per la valutazione della dispnea

#### Grado

- 0 "Mi manca il fiato solo in occasione di attività fisica intensa"
- 1 "Mi manca il fiato se cammino in piano a passo veloce o se percorro una lieve salita a piedi"
- 2 "A causa della mancanza di fiato, cammino in piano più lentamente dei miei coetanei, oppure mi devo fermare per respirare quando cammino in piano al mio passo abituale"
- 3 "Mi devo fermare per respirare dopo aver camminato in piano per circa 100 metri o per pochi minuti"
- 4 "La mia mancanza di fiato è talmente intensa da impedirmi di uscire di casa", o "mi manca il fiato mentre mi vesto"

NB: La scala MRC modificata utilizza gli stessi descrittori della scala MRC originale, nella quale i descrittori sono numerati da 1 a 5. La scala MRC modificata (0-4) è utilizzata per il calcolo dell'indice BODE.

#### - English version

| Table 2.5. Modified MRC dyspnea scale PLEASE TICK IN THE BOX THAT APPLIES TO YOU (ONE BOX ONLY) (Grades 0-4) | |
|---|---|
| mMRC Grade 0. I only get breathless with strenuous exercise. | ۵ |
| mMRC Grade 1. I get short of breath when hurrying on the level or walking up a slight hill. | ٥ |
| mMRC Grade 2. I walk slower than people of the same age on the level because of breathlessness, or I have to stop for breath when walking on my own pace on the level. | 0 |
| mMRC Grade 3. I stop for breath after walking about 100 meters or after a few minutes on the level. | |
| mMRC Grade 4. I am too breathless to leave the house or I am breathless when dressing or undressing. | |

<sup>&</sup>lt;sup>a</sup> Fletcher CM. BMJ 1960; 2: 1662.

#### 8.3 Treatment Satisfaction Questionnaire for Medication (TSQM-9)

- Italian version (used in the SAT study)

# TSQM-9 (italiano)

#### Questionario sulla soddisfazione riguardo al farmaco

Istruzioni – Rifletta sul suo livello di soddisfazione o insoddisfazione riguardo al farmaco che le viene prescritto in questa sperimentazione clinica. Vorremmo la sua opinione sull'efficacia, gli effetti collaterali e la praticità del farmaco durante le ultime 2-3 settimane o dall'ultima volta che lo ha usato. Per ogni domanda, contrassegni solo la risposta che meglio corrisponde alle sue esperienze.

| disfatto/a della capacità del farmaco di prevenire o trattare il suo |
|----------------------------------------------------------------------|
| √a |
| 'a |
| disfatto/a del modo in cui il farmaco allevia i suoi sintomi? |
| √a |
| a |
| disfatto/a del tempo che il farmaco impiega ad agire? |
| /a |
| /a |
| piego del farmaco nella sua forma attuale? |

| 5. Q | uanto è facile o difficile pianificare quando usare il farmaco ogni volta? |
|---|---|
| П. | Estremamente difficile |
| _000 | Molto difficile |
| 1000 | Difficile |
| 0.00 | Relativamente facile |
| | Facile |
| Company of the last | Molto facile |
| 7.00 | Estremamente facile |
| 6. Q | uanto è comodo o scomodo seguire le istruzioni per l'impiego del farmaco? |
| $\Box_1$ | Estremamente scomodo |
| $\square_2$ | Molto scomodo |
| $\square_3$ | Scomodo |
| $\square_4$ | Relativamente comodo |
| $\square_5$ | Comodo |
| $\Box_6$ | Molto comodo |
| $\square_7$ | Estremamente comodo |
| 7. Co | omplessivamente, quanto è sicuro/a che il farmaco le sia di giovamento? |
| $\Box_1$ | Per niente sicuro/a |
| $\square_2$ | Poco sicuro/a |
| $\square_3$ | Abbastanza sicuro/a |
| $\square_4$ | Molto sicuro/a |
| $\square_5$ | Estremamente sicuro/a |
| 8. Q | uanto è sicuro/a che i vantaggi offerti dal farmaco superino gli svantaggi? |
| 200 | Per niente sicuro/a |
| | Poco sicuro/a |
| 100 | Abbastanza sicuro/a |
| | Molto sicuro/a |
| $\sqcup_5$ | Estremamente sicuro/a |
| 9. Tı | atto considerato, quanto è soddisfatto/a o insoddisfatto/a del farmaco? |
| | Estremamente insoddisfatto/a |
| - | Molto insoddisfatto/a |
| | Insoddisfatto/a |
| 2 ( ** | Moderatamente soddisfatto/a |
| - | Soddisfatto/a |
| | Molto soddisfatto/a |
| $\square_7$ | Estremamente soddisfatto/a |

- English version

# TSQM-9

Abbreviated Treatment Satisfaction Questionnaire for Medication

Instructions: Please take some time to think about your level of satisfaction or dissatisfaction with the medication you are taking in this clinical trial. We are interested in your evaluation of the effectiveness, side effects, and convenience of the medication over the last two to three weeks, or since you last used it. For each question, please place a single check mark next to the response that most closely corresponds to your own experiences.

| 1. H | ow satisfied or dissatisfied are you with the ability of the medication to prevent or treat your condition? |
|---|---|
| $\square_1$ | Extremely Dissatisfied |
| $\square_2$ | Very Dissatisfied |
| $\square_3$ | Dissatisfied |
| $\square_4$ | Somewhat Satisfied |
| $\square_5$ | Satisfied |
| $\square_6$ | Very Satisfied |
| $\square_7$ | Extremely Satisfied |
| 2. H | ow satisfied or dissatisfied are you with the way the medication relieves your symptoms? |
| $\square_1$ | Extremely Dissatisfied |
| $\square_2$ | Very Dissatisfied |
| $\square_3$ | Dissatisfied |
| $\square_4$ | Somewhat Satisfied |
| $\square_5$ | Satisfied |
| $\square_6$ | Very Satisfied |
| $\square_7$ | Extremely Satisfied |
| 3. H | ow satisfied or dissatisfied are you with the amount of time it takes the medication to start working? |
| | Extremely Dissatisfied |
| $\square_2$ | Very Dissatisfied |
| | Dissatisfied |
| $\square_4$ | Somewhat Satisfied |
| $\square_5$ | Satisfied |
| $\square_6$ | Very Satisfied |
| $\square_7$ | Extremely Satisfied |
| 4 77 | |
| | ow easy or difficult is it to use the medication in its current form? |
| | Extremely Difficult |
| | Very Difficult |
| _ ` | Difficult |
| $\bigsqcup_4$ | Somewhat Easy |
| _ ` | Easy |
| | Very Easy |
| Ш7 | Extremely Easy |

5. How easy or difficult is it to plan when you will use the medication each time?

| $ \Box_2 $ $ \Box_3 $ $ \Box_4 $ $ \Box_5 $ $ \Box_6 $ | Extremely Difficult Very Difficult Difficult Somewhat Easy Easy Very Easy Extremely Easy |
|---|---|
| | ow convenient or inconvenient is it to take the medication as instructed? |
| | Extremely Inconvenient |
| | Very Inconvenient |
| | Inconvenient |
| | Somewhat Convenient |
| | Convenient |
| | Very Convenient |
| $\sqcup_7$ | Extremely Convenient |
| 7. Ov | verall, how confident are you that taking this medication is a good thing for you? |
| | Not at All Confident |
| | A Little Confident |
| $\square_3$ | Somewhat Confident |
| $\square_4$ | Very Confident |
| $\square_5$ | Extremely Confident |
| | ow certain are you that the good things about your medication outweigh the bad things? |
| | Not at All Certain |
| | A Little Certain |
| _ | Somewhat Certain |
| _ | Very Certain |
| $\bigsqcup_5$ | Extremely Certain |
| 9. Ta | iking all things into account, how satisfied or dissatisfied are you with this medication? |
| $\square_1$ | Extremely Dissatisfied |
| $\square_2$ | Very Dissatisfied |
| $\square_3$ | Dissatisfied |
| $\square_4$ | Somewhat Satisfied |
| $\square_5$ | Satisfied |
| $\Box_6$ | Very Satisfied |
| $\square_7$ | Extremely Satisfied |

#### 8.4 COPD Assessment Test (CAT)

- Italian version (used in the SAT study)

| Nome: | Data di oggi: | CAT |
|-------|---------------|----------------------|
| | | COPD Assessment Test |

# Come va la Sua broncopneumopatia cronica ostruttiva (BPCO)? Esegua il COPD Assessment Test™ (test di valutazione della BPCO) (CAT)

Questo questionario denominato CAT - COPD Assessment Test™ (che significa test per la valutazione della (BPCO)), aiuterà sia Lei che l'operatore sanitario a misurare l'impatto della BPCO sul Suo benessere e sulla Sua vita quotidiana. Le Sue risposte e punteggi del test possono essere utilizzati sia da Lei che dall'operatore sanitario per migliorare la gestione della Sua BPCO e per ottenere i massimi vantaggi dal trattamento.

| | di seguito, inserisca un segno (X) nell<br>re solo una risposta per ogni domano | |
|---|---|---|
| Esempio: Sono molto contento | 0 (2 3 4 5) | Sono molto triste PUNTEGGI |
| Non tossisco mai | 012345 | Tossisco sempre |
| Il mio petto è<br>completamente libero da<br>catarro (muco) | 012345 | Il mio petto è tutto pieno di catarro (muco) |
| Non avverto alcuna sensazione di costrizione al petto | 012345 | Avverto una forte sensazione di costrizione al petto |
| Quando cammino in salita o<br>salgo una rampa di scale non<br>avverto mancanza di flato | 012345 | Quando cammino in salita o<br>salgo una rampa di scale<br>avverto una forte mancanza<br>di flato |
| Non avverto limitazioni<br>nello svolgere qualsiasi<br>attività in casa | 012345 | Avverto gravi limitazioni<br>nello svolgere qualsiasi<br>attività in casa |
| Mi sento tranquillo ad<br>uscire di casa nonostante la<br>mia maiattia polmonare | 012345 | Non mi sento affatto<br>tranquillo ad uscire di casa a<br>causa della mia malattia<br>polmonare |
| Dormo profondamente | 012345 | Non riesco a dormire<br>profondamente a causa della<br>mia maiattia polmonare |
| Ho molta energia | 012345 | Non ho nessuna energia |
| II logo COPD Assessment Test e CAT è i<br>© 2009 GlaxoSmithKline group of compa<br>Last Updated: February 26, 2012 | un marchio registrato del gruppo di società Glaxo<br>unies. Tutti i diritti riservati. | pSmithKline. PUNTEGGIO TOTALE |

# - English version

| | | | TAT |
|---|---|---|---|
| Your name: | | <u>&gt;</u> | |
| Today's date: | | COPD | Assessment Test |
| (Chronic Obstructive Pulmonary<br>answers, and test score, can be<br>the management of your COPE | and your healthcare profess<br>y Disease) is having on your<br>e used by you and your healt<br>and get the greatest benefit<br>back (X) in the box that best d<br>ach question. | ional measure the impact COPE<br>wellbeing and daily life. Your<br>hcare professional to help impro | ve |
| | | | SCORE |
| I never cough | 0 1 2 3 4 9 | I cough all the time | |
| I have no phlegm (mucus)<br>in my chest at all | 0 1 2 3 4 5 | My chest is completely full of phlegm (mucus) | |
| My chest does not feel tight at all | 0 1 2 3 4 5 | My chest feels very tight | |
| When I walk up a hill or one flight of stairs I am not breathless | 0 1 2 3 4 5 | When I walk up a hill or one flight of stairs I am very breathless | |
| I am not limited doing any activities at home | 0 1 2 3 4 3 | I am very limited doing activities at home | |
| I am confident leaving my<br>home despite my lung<br>condition | 0 1 2 3 4 5 | I am not at all confident<br>leaving my home because of<br>my lung condition | |
| I sleep soundly | 0 1 2 3 4 5 | I don't sleep soundly<br>because of my lung condition | |
| I have lots of energy | 0 1 2 3 4 9 | I have no energy at all | |
| COPD Assessment Test and © 2009 GlaxoSmithKline. All | the CAT logo are trademarks of the rights reserved. | TOTAL SCORE GlaxoSmithKline group of companies. | |

MOD 1037.B Rev 01 del 15-11-2012 modified on 1st April 2016

# 8.5 Brief Illness Perception Questionnaire (B-IPQ)

- Italian version (used in the SAT study)

Per le seguenti domande, per favore cerchi il numero che meglio corrisponde al suo punto di vista.

| Quanto la su | a mala | ttia in | fluenza | la sua v | vita? | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Non l'influen | 1<br>za per r | 2<br>nulla | 3 | 4 | 5 | 6 | 7 | 8 | 9<br>la infl | 10<br>luenza gravemente |
| Per quanto t | empo p | ensa l | a sua m | alattia | continu | uerà? | | | | |
| Per un tempo | 1<br>molto l | 2<br>breve | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>per sempre |
| Quanto cont | rollo cr | ede di | avere | sulla su | a malat | ttia? | | | | |
| Assolutament<br>controllo | 1<br>e nessu | 2<br>in | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>un controllo<br>assoluto |
| Quanto pens | a che il | suo ti | attame | nto (pil | lole, ec | c.) pos | s <mark>a ai</mark> uta | are la s | ua mal | attia? |
| Per nulla | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9<br>Estre | 10<br>mamente di aiuto |
| Quanto sente | i sinto | mi de | lla sua i | malattia | a? | | | | | |
| Alcun sintom | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9<br>Sinto | 10<br>mi molto gravi |
| Quanto è pre | occupa | ito pei | la sua | malatti | a? | | | | | |
| Per nulla prec | 1<br>occupate | 2 | 3 | 4 | 5 | 6 | 7 | 8<br>Estre | 9<br>emamen | 10<br>te preoccupato |
| Quanto cred | e di cap | pire be | ne la su | ıa mala | ttia? | | | | | |
| Per nulla | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9<br>Capit | 10<br>a molto chiaramente |
| Quanto la su<br>turbare, dep | | | na cam | biato le | sue e | mozion | i? (ad | es. la | fa arra | bbiare, spaventare |
| Non ha camb | | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | 10<br>nbiato estremamente<br>ozioni |
| Per favore, e<br>malattia: | lenchi i | in ord | ine di ir | nportai | nza i tro | e fattor | i princ | ipali cl | he hann | o causato la sua |

# - English version

#### The Brief Illness Perception Questionnaire

For the following questions, please circle the number that best corresponds to your views:

| How muc | h does | your il | lness a | ffect y | our life | ? | | 8132 | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 0<br>no affect<br>at all | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>severely<br>affects my life |
| How long | How long do you think your illness will continue? | | | | | | | | | |
| 0<br>a very<br>short time | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>forever |
| How much control do you feel you have over your illness? | | | | | | | | | | |
| 0<br>absolutely<br>no control | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>extreme amount<br>of control |
| How muc | h do yo | u thin | your f | treatme | nt can | help yo | ur illne | ess? | | |
| 0<br>not at all | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>extremely<br>helpful |
| How muc | h do yo | ou expe | rience | sympt | oms fro | m you | illnes | s? | | |
| 0<br>no sympto<br>at all | 1<br>ms | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>many severe<br>symptoms |
| How cond | erned | are you | ı about | your il | Iness? | | | | | |
| 0<br>not at all<br>concerned | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>extremely<br>concerned |
| How well | do you | feel yo | ou und | erstand | l your il | Iness? | | | | |
| 0<br>don't unde<br>at all | 1<br>rstand | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>understand<br>very clearly |
| How muc<br>upset or o | | | lness a | iffect ye | ou emo | tionally | /? (e.g. | does it | t make | you angry, scared, |
| 0<br>not at all<br>affected<br>emotionall | 1<br>y | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>extremely<br>affected<br>emotionally |
| Please lis<br>illness. Ti<br>1<br>2 | t in ran<br>ne mos | t impoi | rtant ca | | or me:- | ortant fa | actors | that yo | u believ | ve caused <u>vour</u> |

@ All rights reserved. For permission to use the scale please contact:

# 8.6 Morisky Medication Adherence Scale (MMAS-4)

- Italian version (used in the SAT study)

# **Morisky Medication Adherence Scale (©MMAS-4)**

| Le capita mai di dimenticarsi di prendere i suoi farmaci per la BPCO? | Sì<br>□ | No<br>□ | |
|---|---|---|---|
| 2*. Le capita mai di avere problemi a ricordarsi di prendere i suoi farmaci per la BPCO? | | ٠ | |
| 3. Quando si sente meglio, a volte smette di prendere i suoi farmaci per la BPCO? | | ۵ | |
| 4. Se a volte si sente peggio quando prende i suoi farmaci per la BPCO, smette di prenderli? | | ٥ | |
| - English version Morisky Medication Adherence Scale (©MMAS-4) | | | |
| (Please check one box on each line) | | | - |
| Do you ever forget to take your (name of health condition) medicine? | Yes<br>□ | No<br>□ | |
| 2*. Do you ever have problems remembering to take your (name of health condition) medication? | | ٠ | |
| 3. When you feel better, do you sometimes stop taking your (name of health condition) medicine? | | ٥ | |
| <ul> <li>4. Sometimes if you feel worse when you take your (name of health condition) medicine, do you stop taking it?</li> <li>*modified item from original scale appearing in Medical Care 1986</li> </ul> | | ۵ | |